### GT Biopharma, Inc.

# GTB-3550 (CD16/IL-15/CD33) Tri-Specific Killer Engager (TriKE™) for the Treatment of High Risk Myelodysplastic Syndromes, Refractory/Relapsed Acute Myeloid Leukemia and Advanced Systemic Mastocytosis

### **IND Sponsor:**

GT BIOPHARMA, INC. 9350 Wilshire Blvd Suite 203 Beverly Hills, CA 90212

Version Date:
June 4, 2021 / Revision 13
Confidential

# **Key Study Personnel Contact Information**



Refer to the Procedures Manual for Participating Sites for a complete list of study personnel and contact information.

June 4, 2021 

# **Revision History**

| Revision | Version | Summary of Changes | Consent |
|---|---|---|---|
| # | Date<br>12/28/2016 | Original to CRRC | Changes |
| | 02/16/2017 | Original to CPRC In response to CPRC stipulations: | n/a |
| | 02/10/2017 | Delete CML from inclusion and CML in blast crisis from exclusion | |
| | | Add inclusion criteria for ALL | |
| | 05/19/2017 | <ul> <li>In response to CPRC stipulations, original version to FDA</li> <li>Study Schema, Page 8 – Correct to reflect that early study stopping rules only apply to the extended cohort</li> <li>Synopsis, Section 5.1, Appendix 1 – further define advanced systemic mastocytosis</li> <li>Other edits based FDA's comments as part of the pre-IND and general</li> </ul> | n/a |
| | | <ul> <li>edits:</li> <li>Clarify dose escalation component is done as inpatient, extended component may be as an outpatient after the 1<sup>st</sup> 24 hours</li> <li>Add upper age limit of 75 years</li> <li>Section 8.2 add overview of correlative testing</li> <li>Clarify CD33 testing for eligibility will be by flow cytometry or IHC</li> <li>Clarify that dose limiting toxicity is for treatment related events occurring within 28 days of the 1<sup>st</sup> dose and that CRS toxicity uses a modified grading system based on Lee, et al. (otherwise CTCAE v4 is used)</li> <li>Include toxicity profile for blinatumomab as a similar monoclonial antibody since 161533 TriKE has not be tested in humans</li> <li>Updated eligibility to tighten liver function requirements based on experience with DT2219</li> <li>Other minor edits</li> </ul> | |
| | 08/11/2017 | Version submitted to FDA in Serial 001 Updated disease-specific eligibility criteria to clearly exclude patients with good standard of care treatment options Require both patients per dose cohort to complete the DLT evaluation period prior to dose escalation Add pulmonary function testing to eligibility criteria Revised DLT based on FDA guidance Add blood pressure criterion for continuing therapy from Block 2 to Block 3 Clarify that meeting either stopping rule criterion would stop the study. Require that all patients be treated inpatient or on hospital-based Phase I Unit. Add serum pregnancy test within for females of child-bearing potential Fix discrepancy about LFT monitoring for dose adjustments Add serum magnesium and phosphorous evaluations to the Schedule of Assessments Added information about dose preparation and delivery | |
| | 04/23/2018 | In response to FDA request dated 8/23/2017: Exclude diagnosis of acute lymphoblastic leukemia (ALL) Exclude "other CD33 expressing diseases" Update title to reflect above changes Update eligibility to CD33 expressing malignancies, not requiring testing of CD33 status for individual patients Require all treatment to be administered as an inpatient Clarify during phase I 1 patient within a cohort must reach day 28 between enrollment may begin in the next 2 patient cohort Update and clarify definition of dose limiting toxicity Add monitoring for signs of immune activation for all phase I patients and impact plan on future dose level escalation Add monitoring for signs of immune activation for all patients and impact plan on future enrollees | yes |

| Revision<br># | Version<br>Date | Summary of Changes | Consent<br>Changes |
|---|---|---|---|
| | | <ul> <li>Eligibility for PFT's ≥ 80% per FDA</li> <li>Eligibility for LVEF ≥ 45% to match transplant protocols, previously ≥ 40%</li> <li>Add to exclusion criteria "eligible for standard of care transplant"</li> <li>Expand management section for increased LFTs</li> <li>Add management section for pulmonary toxicity</li> <li>Update Section 9 to reflect CMC and product SOPs</li> <li>Update appendices to match protocol changes.</li> </ul> Other protocol revisions: | |
| | | <ul> <li>For AML patients having previous transplant, change key timeframe for eligibility from 12 months to 3 months</li> <li>Update MDS eligibility and add Appendix III IPSS tables and link to calculator</li> <li>TriKE dose dosing units changed to microgram/kg/day (previously mcg/m2) and change dose levels to be tested</li> <li>Remove bolus test dose for phase I patients, move PK/PD sampling until after the end of each block (96 hours or earlier if infusion is ended</li> </ul> | |
| | | <ul> <li>until after the end of each block (96 hours of earlier it infusion is ended earlier) and do for all patients (not just Phase I), updated definition of DLT to remove unable to tolerate bolus dose</li> <li>Change from CTCAE v4 to CTCAE v5</li> <li>Clarify in the primary endpoint for Phase II that response is based on the "best" clinical response by Day 42</li> <li>Section 7.4 Permit retreatment for patients with clinical benefit defined</li> </ul> | |
| | | as stable or better at time of 1 <sup>st</sup> disease reassessment Add additional agent administration info in Section 7.1 Move criteria to begin Block 2 and 3 to Section 7.1 and clarify when to delay start of a new block Define neurologic assessment in Section 7.3.4 Revised research sample table to reflect changes in the protocol | |
| | | <ul> <li>(primarily delete bolus test dose in phase I and move PK/PD sampling to end of block dosing)</li> <li>Update Section 9.7 Potential Toxicities</li> <li>Expand language regarding targeted toxicity and research sample collection if a patient is not continuing study treatment as planned</li> <li>Update MT number to HM</li> </ul> | |
| | | Update cover page and page 3 listing as PI and GT Biopharma as IND Sponsor Other minor edits and clarifications Updates based on surrent protect template: | |
| | | Updates based on current protocol template: Add Key abbreviations table Section 5 patient enrollment updated Update Section 10.1 definitions for event reporting Other minor edits and clarifications | |
| | 07/05/2018 | <ul> <li>In response to FDA's clinical information request dated July 3, 2018</li> <li>Synopsis and including Sections 7.2.1, 12.1 - During dose finding component require both patients reach Day 28 (end of the DLT assessment period) before enrollment of a new cohort – remove reference to time-to-event (TITE) for the continuous reassessment method (CRM) as not long applicable</li> <li>Synopsis, Section 5, Appendix I - Clarify eligibility for relapsed AML in regards to transplant status</li> </ul> | n/a |
| | | <ul> <li>Schema, Sections 7.2.1, 10.2 - Expand general definition of DLT as emergent toxicity with the exception of those that are clearly and incontrovertibly due to extraneous causes</li> <li>Schema, Section 7.2.1, 10.2 - For Grade 3 exceptions add that electrolyte disturbance must resolve, with or without intervention, to &lt;</li> </ul> | |

| Revision<br># | Version<br>Date | Summary of Changes | Consent<br>Changes |
|---|---|---|---|
| " | | Grade 2 levels within 72 hours to not be a DLT, delete skin rash from the list of Grade 3 exceptions Section 7.2, 12.4 - Modify the monitoring period for the early study stopping rule event for Grade 4-5 toxicity from 14 days after the start of the last treatment block to 42 days after the start of the first treatment block Section 5.3, Appendix I – expand exclusion to include a candidate for potentially curative therapy to no previous HSCT exclusion Section 7.1 expand criteria to continue to Block 2 and 3 to include requirements for hem, renal and liver function, adjust criteria to O2 saturation rate to match CTCAE v5 (links to management of pulmonary toxicity Section 7.3.5) Section 7.3.5 – expand management of pulmonary toxicity Section 9.6 – indicate the albumin used in the infusion prep is the commercially available Flexbumin 25% Other edits/clarifications Update abbreviation table to remove TITE Schema, Sections 7.2.1, 10.2 - Definition of DLT "add despite "support with transfusions" to definition for platelet count decreased Section 9 - add general supportive care statement Schema, Sections 7.2.1, 10.2 - Clarify in DLT definition that persons with increased LFT's that met criteria for further treatment in Section 7.3.3 may continue on treatment (in general a DLT in any patient = off | - Thursday |
| | | <ul> <li>7.3.3 may continue on treatment (in general a DLT in any patient = off treatment)</li> <li>Section 7.4 Expand re-treatment and add new Section 8.3 Retreatment Research Related Samples</li> <li>Section 7.1 – clarify a treatment delay of 1 week is permitted (previous language of up to 1 week was unclear)</li> <li>Other minor edits – all tracked in tracked version</li> </ul> | |
| | 07/09/2018 | In response to FDA's 2 <sup>nd</sup> request Synopsis, Section 5.1 and Appendix I – delete AML eligibility criteria permitting enrollment of patients between 3 and 12 most post-transplant Schema, Sections 7.2.1 and 10.2 - delete "despite support with transfusions" from the decreased platelet definition of dose limiting toxicity from synopsis | n/a |
| | | Additional revision: Schema, Sections 7.2.1 and 10.2 - remove febrile neutropenia from the definition of DLT for MDS/Mast cell disorders Update Appendix I exclusion criteria #13 to match previous edit in Section 5.3 | |
| | 10/15/2018 | In response to the FDA's Full Clinical Hold letter received September 28, 2018 (add collection of TriKE samples pre- and post-infusion for batch analysis of drug concentration levels) • Section 7.1 – add instructions for the collection of the post-infusion TriKE sample • Section 8.2 – add drug sample collection pre- and post-infusion to table of research related testing, assessment and sample collection • Section 8.4 – indicate in #5 that the samples will be stored frozen at ≥ 80°F in the Translational Therapy Lab until batch analysis • Section 9.6 – add a bullet point to the drug preparation instructions to collect samples of the final product before the prepared drug leaves the investigational drug services (IDS) pharmacy. In response to the FDA's clinical non-hold issues received July 12, 2018: • Sections 5.2 and 7.4, Appendix I – change eligibility threshold for renal function by eGFR from ≥40 to ≥ 60 mL/min/1.73 m² and change total bilirubin from ≤2.5 mg/dl to ≤ 1.5 x ULN | |

June 4, 2021 

| Revision<br># | Version<br>Date | Summary of Changes | Consent<br>Changes |
|---|---|---|---|
| | | Section 5.3 Exclusion criteria and Appendix I - add exclusions of A family history of long QT syndrome or with a QTc interval > 480 msec at screening AND Currently taking medications known to prolong QT/QTc interval as the potential risk of QT/QTc prolongation is unknown in humans (refer to Appendix VII for a list of prohibited medications for eligibility) | |
| | | <ul> <li>Section 7.3 add a paragraph regarding the use of medications that prolong QT/QTc during the study.</li> <li>Insert a new Appendix VII - Combined List of Drugs That Prolong QT/QTc.</li> </ul> | |
| | | <ul> <li>Sections 7.1 and 7.3 – add language regarding the interactions between TriKE and the P450 system are unknown. And that the IL-15 component may affect the 3A4 and 2D6 substrates. Patients with unexpected toxicity should have a review of their con-meds to determine whether there are any potential interactions. The PI or treating physician should consider discontinuing these medications as clinically indicated.</li> <li>Insert a new Appendix VI – P450 Drug Interactions</li> </ul> | |
| | | <ul> <li>Section 8.1 Required Standard of Care – add collection of concomitant<br/>medications beginning at screen through the end of treatment visit with<br/>start and stop dates relative to TriKE infusions AND ECG at baseline per<br/>Section 5.3 exclusion criteria</li> </ul> | |
| | | <ul> <li>Section 8.2 add antibody testing on Day 15 pre-dosing (using a portion<br/>of the red top tube already being collected at the time point<br/>In response to the continuing clinical hold:</li> </ul> | |
| | | <ul> <li>Update Section 9 161533 TriKE Description, Supply, Preparation based<br/>on pre-clinical function/microbial testing<br/>Other edits and clarifications:</li> </ul> | |
| | | <ul> <li>Remove from cover page as leaving the institution</li> <li>Add as a co-I</li> <li>Add re-treatment enrollment Section 6.4 and a new re-treatment eligibility checklist as Appendix II, Renumber all subsequent appendices</li> <li>Section 8.2 - Reduce the intensity of research sample collection from daily during each TriKE block to prior to a block start and the 3<sup>rd</sup> day of each block with a +2 day window</li> </ul> | |
| | | <ul> <li>Section 8.3 – limit research related sample collection to Block 1 only, while retaining baseline and Day 22 samples</li> <li>Other edits and clarifications detailed in separate summary of revisions log</li> </ul> | |
| 1 | 02/11/2019 | Section 9.2 Product Manufacturing and Section 9.5 Storage and Stability update to match current MCT process with the final product stored in a <-70° C freezer that is locked with limited access Section 8.4 Overview of Planned Correlative – update to <-70° C freezer for research sample storage | Yes – PI<br>name/<br>contact<br>info |
| | | Cover page, contact information, Replace as PI with (currently a co-I) as is leaving UMN Synopsis, Section 5.1, Appendices I and IV - Delete references to old IPSS MDS criteria (study already uses R-IPSS) | |
| | | <ul> <li>Appendix V - Add hematologic improvement criteria to MDS response criteria</li> <li>Section 8.3 Re-Treatment Research samples – edit the Block 1 header to eliminate stray words</li> </ul> | |
| 2 | 07/26/2019 | Updated version based on teleconference July 26, 2019 Section 8.2 – Add daily a EKG to collect additional safety data during each of the 3 blocks of treatment at 4 hours (±15 minutes) into the each infusion start and at 4 hours (±15 minutes) after the infusion disconnection on the last day of the block Section 10.3 – update MCC required reporting to IND Sponsor | yes |

| Revision<br># | Version<br>Date | Summary of Changes | Consent<br>Changes |
|---|---|---|---|
| | | <ul> <li>Renumber references deleting references removed in July 2018 revision</li> <li>Previous edits July 10, 2019 version Based on SIV:</li> <li>Section 5.3, Appendices 1 and 2: clarify HIV status as "known history of HIV"</li> <li>Section 7.1 and Section 7.3.2: replace references to hypersensitivity and allergic/anaphylactic with infusion related reaction as the study switched to CTCAE v 5 in the April 2018 protocol version – makes consistent with DLT definition and Appendix VIII Targeted Toxicity Worksheet use of infusion related reaction</li> <li>Synopsis, Section 4 and Section 10.2 Update wording on Dose Limiting Toxicities (DLT) to</li> <li>Resolve discrepancies in wording found in the protocol and to clarify hematologic parameters for toxicity given the baseline hematologic abnormalities inherent to AML and MDS:</li> <li>Updated hematologic toxicity parameters as the standard grading system does not apply to AML and MDS patients given their baseline platelets/neutrophils already meet grade 3 and 4 due to the disease process itself.</li> <li>Added Grade 3 Infection to the exclusions for DLT given that infection is inherent in MDS/AML as a disease related complication</li> <li>Section 9.6, 5th bullet final product samples: delete the words "to be handed to the infusion team member along with the infusion bag and tubing" to make consistent with rest of language in bullet and Section</li> </ul> | |
| | | 8.2 as left over wording from a previous revision Updated Appendix I and II to new CTO format for eligibility checklists | |
| 3 | 09/23/2019 | Throughout protocol: Replace the product name 161533 TriKEs with GTB-3550 TriKE™ Appendices I and II: Delete Eligibility Checklists per new CTO policy and renumber remaining appendices | Update<br>product<br>name |
| 4 | 12/18/2019 | <ul> <li>The following changes are made to the inclusion/exclusion criteria:</li> <li>Synopsis and Section 5.1: Patients with AML who relapse 3 months after transplant may be included only if off immunosuppression for a minimum of 4 weeks and do not have GVHD. Rationale: Patients who relapse after transplant have no other good therapeutic options.</li> <li>Section 5.2: Remove upper age limit. Rationale: Avoids exclusion of older patients who otherwise would be eligible for study participation.</li> <li>Section 5.2: Redefine the pulmonary function as DLCO corrected (ml/min/mm Hg) as no more than 5 units below lower limit of normal (CTCAE v5 Grade 1 carbon monoxide diffusing capacity decreased) based on patient's height, weight, and gender as reported by the institutional pulmonary function lab.</li> <li>The following changes reflect moving from a single center study to multisite study</li> <li>Throughout protocol: Update the study to include participating sites template language.</li> <li>Update protocol to reflect external monitoring by GT Biopharma or designee for all sites.</li> <li>Other protocol revision:</li> <li>Section 12.4 – Expand actions associated with an early stopping rule event to allow a temporary halt of enrollment while reviewing the event rather than stopping the study.</li> <li>Clarifications:</li> <li>Section 7.1 post-infusion TriKE product collection – revise to allow sample collection either on the unit or in the institutional research lab</li> </ul> | Yes |

| Revision<br># | Version<br>Date | Summary of Changes | Consent<br>Changes |
|---|---|---|---|
| | | Section 7.3 – add a reminder any patient experiencing a DLT equivalent toxicity must discontinue therapy and is not eligible for retreatment Section 10.2 – clarify event monitoring begins with the 1st dose of TriKE | |
| 5 | 01/30/2020 | Section 5.3 – Change driving time requirement from 45 minutes to 90 minutes | No |
| 6 | 02/12/2020 | Section 5.2 – Change "and" to "or": Absolute lymphocyte count (ALC) $\geq$ 200 cells/mm³ OR absolute circulating CD56+/CD3- NK cell count >25 cells/µL within the 14 days prior to start of therapy. Rationale: More precise characterization of goal to maximize NK cells as the primary cell of interest and mechanism of action ( MOA) | No |
| 7 | 04/10/2020 | Section 7.4 and Section 8 – add language to clarify that the standard of care procedures in Section 8.1 should be followed for patients who are enrolled for retreatment. Section 8.1 – clarified timing of procedures on the days of infusion. Consent changes – added background information to retreatment consent and updated long term specimen storage language to state that samples will be under the control of GT BioPharma. | Yes |
| 8 | 05/18/2020 | Study Schema, Section 7.2, and Section 10.3 –DLT assessments are protocol defined at Day 29. We recognized that our currently approved protocol has 2 different dates for assessment in the DLT section (Day 29 for non-hematologic and Day 42 for Hematologic assessment) which is incongruent. Thus, revised DLT assessments to clarify that hematological toxicity will be defined as lasting ≥ 29 days from start of cycle as all DLT assessments need to have the same timeline to be congruent with moving forward with subsequent patients at 29 days. | No |
| 9 | 08/31/2020 | Section 7.1.5 and Section 7.5 – clarify that if after completing Block 1 and Block 2 patients with clear evidence of disease progression will discontinue treatment but will be fully evaluable for toxicity and efficacy Section 7.1 and Section 9.6 – Update the drug preparation instructions to match the study's Pharmacy Manual Section 12. 1 – add the definition of evaluable and when to replace a patient to complete enrollment. Other minor edits and clarifications | No |
| 10 | 10/05/2020 | Synopsis, Section 6.4 and Section 7.4 - clarify when re-treatment may be considered. Section 10.6 – Delete from the list of persons who receive participating sites event reports for initial review. Section 10.7 – Clarify UMN's reporting flow to GTB and for SAEs, remove link for MCC SAE reporting as process has changed and receiving report notification via Section 11.3 – Clarify that this study complies with the Masonic Cancer Data and Safety Monitoring Plan (DSMP) and add the link to the plan. Section 11.5 – add ICH compliant record retention information. Other minor edits and clarifications. | No |
| 11 | 03/25/2021 | Section 5.1 - updated definition of CD33-expressing myeloid malignancies to include phrase with greater than or equal to 50% CD33+ target cells in order to maximize potential patient benefit of treatment with GTB-3550 Added new eligibility for Elderly AML not fit for induction therapy can be enrolled after 2 failed inductions Section 5.2 updated ranges for hepatic function in order to limit pre-existing liver abnormalities Section 5.3 added new exclusions to reduce risk of comorbidities; concomitant active cancer, severe clinical obesity, over-the counter medication. Added new Section 6.2 Prior and Concomitant Therapy in order to document the review of the non-study medication used by the patient by both the Investigator and GT Biopharma. | No |

June 4, 2021 

| Revision<br># | Version<br>Date | Summary of Changes | Consent<br>Changes |
|---|---|---|---|
| | | Section 7.1.3 Supportive Care/Concomitant Medications added language regarding potential risk of LFT elevations. To reduce the risk of comorbidities, the use of medications known to elevate LFTs are prohibited from screening and the end of treatment visit. Section 7.2.1 DLT clarified the use of LFT results. Section 7.3.3 updated management of abnormal LFT results to enhance patient safety by stipulating a longer recovery time. Section 8.1 added INR testing to screening labs; added abdomen scan to CTs to allow for review of liver abnormalities and pre-existing conditions. Section 10.3 excluded grade 3 LFTs from DLT list Section 10.4 and section 10.5 clarified sponsor responsibility. | |
| 12 | 05/07/2021 | Section 7.2.1 Corrected language under Additional Dose Escalation Parameters. Rationale: This revision is to resolve an error (and inconsistency) in the written protocol. The intent of this statement was based on FDA comments to proceed more cautiously than dose doubling if we started to see signs of immune activation. Schema, Section 7.2.1 Added new dose level at 150 mcg/kg/day. Rationale, to slow down dose escalation when immune activation is possible, rather than proceeding from 100 mcg/kg/day to 200 mcg/kg/day as written, we will enroll the next cohort at 150 mcg/kg/day. Section 12.1 Updated statistics – rationale to account for new dose level Throughout protocol – updated to note that 7 dose levels are being tested Section 12.1 removed outdated reference to 2 mcg/kg/day – rationale, error correction – study never used this dose level. | Yes |
| 13 | 06/01/2021 | Key Study Personnel – Updated University of Minnesota. Synopsis, Section 7.2.1 and Section 10.3 – Updated DLT language to clarify DLT must be treatment related to GTB-3550 within 28 days as assessed on Day 29 from the first dose. Furthered clarified Grade 3 non-hematologic adverse events lasting more than 72 hours, with the exceptions noted, are DLTs. Added non-sustained Grade 3 QTc in the absence of cardiac arrhythmias (< 72 hours) is not a DLT. Added units to neutrophil and platelet count. Section 9.6 – Added language for paclitaxel non-DEHP equivalent tubing as determined by GTB can be used with GTB-3550 administration. | |

# **Table of Contents**

| Key Abbre | eviations | 13 |
|---|---|---|
| Protocol S | ynopsis | 14 |
| Study Sch | ema | 17 |
| 1 Object | tives | 19 |
| 1.1 F | Primary Objective | 19 |
| 1.2 | Secondary Objectives | 19 |
| 1.3 | Correlative (Research) Objectives | 19 |
| 2 Back | ground | 19 |
| 3 Sumn | nary and Rationale | 21 |
| 4 Study | Design | 22 |
| 5 Patier | nt Selection | 24 |
| | ligible Diseases | |
| | age, Performance Status, Organ Function, Contraception Use | |
| | xclusion Criteria | |
| | nt Screening and Study Enrollment | |
| | Consent and Study Screening in UMN | |
| | Prior and Concomitant Therapy: | |
| | Study Enrollment and GTB-3550 TriKE Dose Level | |
| | nability to Begin Study Treatment | |
| | Re-Treatment Enrollment onto 2015LS167R | |
| | ment Plan | |
| | GTB-3550 TriKE Administration | |
| 7.1.1 | Monitoring Requirements During TriKE Infusions | |
| 7.1.2 | Monitoring for Signs of Immune Activation (Phase I Patients): | |
| 7.1.3 | Supportive Care/Concomitant Medications | 30 |
| 7.1.4 | Dose Modifications. | 31 |
| 7.1.5 | Criteria to Continue with GTB-3550 TriKE Block #2 and #3 | 31 |
| 7.2 | STB-3550 TriKE Dose Levels | 32 |
| 7.2.1 | Dose Finding Component (Phase I) | 32 |
| 7.2.2 | Extended Component (Phase II) | 34 |
| 7.3 N | Management of Selected GTB-3550 TriKE Toxicities | 35 |
| 7.3.1 | Tumor Lysis Syndrome | 35 |
| 7.3.2 | Infusion Related Reaction | 35 |
| 7.3.3 | Increase in Liver Function Tests | 35 |

| | 7.3 | 4 Neurotoxicity | 36 |
|---|---|---|---|
| | 7.3 | .5 Pulmonary Toxicity | 36 |
| | 7.3 | .6 Cytokine Release Syndrome (CRS) or CRS-Like Symptoms | 36 |
| | 7.4 | Opportunity for Re-Treatment | |
| | 7.5 | Duration of Study Treatment | 37 |
| | 7.6 | Duration of Study Participation | 37 |
| 8 | Sch | nedule of Patient Activities | 38 |
| | 8.1 | Required Standard of Care | 39 |
| | 8.2 | Research Related Testing, Assessments, and Sample Collections | 41 |
| | 8.3 | Re-Treatment Research Related Testing, Assessments, and Sample Collections | 43 |
| | 8.4 | Overview of Planned Correlative Studies | 44 |
| 9 | GT | B-3550 TriKE Description, Supply, Preparation, and Potential Toxicities | 45 |
| | 9.1 | Product Description. | 45 |
| | 9.2 | Product Manufacturing | 45 |
| | 9.3 | Product Formulation | 45 |
| | 9.4 | How Supplied | 45 |
| | 9.5 | Study Site Storage and Product Stability | 46 |
| | 9.6 | Preparation and Administration | 46 |
| | 9.7 | Potential Toxicities | 47 |
| 1( | 0 Eve | ent Monitoring, Documentation and Reporting | 48 |
| | 10.1 | Definitions | 48 |
| | 10.2 | Event Documentation | 50 |
| | 10.3 | Dose Limiting Toxicity Documentation and Reporting (Phase I Dose Finding) | 51 |
| | 10.4 | Early Study Stopping Rules - Event Documentation and Reporting (Phase II Dose | 52 |
| | | nsion) Documentation of Death and Reporting Requirements | |
| | 10.5 | Participating Sites Event Reporting Table | |
| | 10.7 | UMN Required Reporting: UMN IRB, GT Biopharma, and Masonic Cancer | 54 |
| | | er's SAE Coordinator, and wasonic Garicer | 54 |
| 1 | 1 Stu | dy Data Collection and Monitoring | 55 |
| | 11.1 | Data Management | 55 |
| | 11.2 | Case Report Forms | 55 |
| | 11.3 | Data and Safety Monitoring | 55 |
| | 11.4 | UMN Led Teleconferences – Participating Sites, GT Biopharma and | 56 |
| | 11.5 | Record Retention | 56 |
| 1: | 2 Sta | tistical Considerations | 57 |
| | 12.1 | Study Design and Endpoints | 57 |

| 12.2 | Statistical Analysis | .59 |
|---|---|---|
| 12.3 | Sample Size Justification | .59 |
| 12.4 | Monitoring Guidelines (Study Stopping Rule Events) | .60 |
| 13 Con | duct of the Study | .61 |
| 13.1 | Good Clinical Practice | .61 |
| 13.2 | Ethical Considerations | .61 |
| 13.3 | Informed Consent | .61 |
| 14 Refe | erences | .62 |
| Appendi | x I - Karnofsky Performance Status | .65 |
| | x II - Revised International Prognostic Scoring System (IPSS-R) for Myelodysplastic nes and Risk Assessment Calculator Link | .66 |
| Appendi | x III - Response Criteria | .68 |
| Appendi | x IV - P450 Drug Interactions | .69 |
| Appendi | x V - Combined List of Drugs That Prolong QT/QTc | .74 |
| ∆nnendi | y VI - Targeted Expected Toxicities Worksheet | 70 |

# **Key Abbreviations**

| antibody-dependent cell-mediated cytotoxicity |
|-------------------------------------------------|
| Adverse event |
| Absolute lymphocyte count |
| Acute myeloid (myelogenous) leukemia |
| chimeric antigen receptor |
| Continuous infusion |
| Central nervous system |
| Complete remission |
| Complete remission with incomplete hem recovery |
| continual reassessment method |
| Complete remission without platelet recovery |
| Cytokine Release Syndrome |
| Common Terminology Criteria for Adverse Events |
| Clinical Trials Office |
| dose limiting toxicity |
| Data and Safety Monitoring Council |
| electronic case report form |
| Food and Drug Administration |
| Graft versus host disease |
| hematologic improvement |
| investigational new drug |
| Revised International Prognostic Scoring System |
| Institutional Review Board |
| Intravenous (into a vein) |
| Laboratory Information Management System |
| monoclonal antibodies |
| Masonic Cancer Center |
| myelodysplastic syndrome |
| myeloid derived suppressor cells |
| maximum tolerated dose |
| natural killer |
| overall survival |
| pulmonary function tests |
| pharmacokinetic/pharmacodynamics |
| per os (by mouth) |
| serious adverse event |
| Tri-Specific Killer Engager |
| Translational Therapy Laboratory |
| University of Minnesota |
| WHO Based Prognostic Scoring System |

#### **Protocol Synopsis**

GTB-3550 (CD16/IL-15/CD33) Tri-Specific Killer Engager (TriKE™) for the Treatment of High Risk Myelodysplastic Syndromes, Refractory/Relapsed Acute Myeloid Leukemia and Advanced Systemic Mastocytosis

# Study Design:

This is a multisite Phase I/II clinical trial of GTB-3550 (CD16/IL-15/CD33) tri-specific killer cell engager (TriKE™) for the treatment of CD33-expressing high-risk myelodysplastic syndromes, refractory/relapsed acute myeloid leukemia or advanced systemic mastocytosis. Up to 10 sites may participate. The hypothesis is that GTB-3550 TriKE will induce natural killer cell function by targeting malignant cells as well as CD33⁺ myeloid derived suppressor cells (MDSC) which contribute to tumor induced immunosuppression. Because CD16 is the most potent activating receptor on NK cells, this single agent may induce a targeted anti-CD33⁺ tumor response.

Patients receive a single course of GTB-3550 TriKE given as 3 weekly treatment blocks. Each block consists of four consecutive 24 hour continuous infusions of GTB-3550 TriKE followed by a 72 hour break after Block #1 and #2. All treatment is given as an inpatient.

Disease response is assessed by bone marrow biopsy performed between Day 21 and Day 42 after the start of the 1<sup>st</sup> infusion. Follow-up for response and survival continues through 6 months from treatment start. Patients experiencing lack of disease progression or evidence of clinical improvement and no unacceptable side effects may be considered for a 2<sup>nd</sup> course of GTB-3550 TriKE on a compassionate basis.

The study consists of two components. The dose finding component is a modified version of a Phase I trial and the extended component is a modified Phase II trial.

#### **Phase I Dose Finding Component:**

The Phase I component uses a continual reassessment method (CRM) to determine the maximum tolerated dose (MTD) of GTB-3550 TriKE. Up to 7 doses levels will be tested. The goal of the CRM is to identify the dose level which most closely corresponds to the targeted dose limiting toxicity (DLT) rate of 20%. Patients are enrolled in cohorts of 2 beginning at Dose Level 1. A minimum of 1 week must separate each patient. Both patients within a cohort must reach Day 28 (end of the DLT assessment period) prior to enrollment of a subsequent cohort. The study statistician assigns each new cohort of 2 patients to the most appropriate dose level based on updated toxicity probabilities. As enrollment proceeds, each cohort is assigned to an increased, decreased or equivalent dose level based on prior data in the trial until the study sample reaches 30. At this time, the last dose is declared the MTD and becomes the GTB-3550 TriKE dose for the extended component.

### **Phase II Extended Component:**

The primary goal of the extended component is to study the potential efficacy of GTB-3550 TriKE in this patient population. Efficacy is measured using rates of complete and partial remission. A Simon's MiniMax two-stage design is used in this phase. Stage 1 will enroll 13 patients, including all patients treated at the MTD defined during the dose finding component. If 3 or more of these 13 patients experience a clinical response by Day 42, the trial moves to Stage 2 and enrolls an additional 17 patients. If at least 10 of the 30 patients have a disease response, GTB-3550 TriKE will be considered for further investigation. There is no staggering of enrollment for this cohort.

# Primary Objectives:

<u>Phase I Dose Finding:</u> To identify the maximum tolerated dose (MTD) of GTB-3550 TriKE defined as the dose level that most closely corresponds to a dose limiting toxicity rate (DLT) of 20%.

<u>Phase II Extension</u>: To determine preliminary efficacy as measured by the rates of "best" clinical response by Day 42 day after the start of the 1<sup>st</sup> infusion. For AML clinical response includes complete remission with or without hematologic or platelet recovery (CR, CRi or CRp) or partial response. For MDS clinical response includes complete remission, marrow CR (with incomplete peripheral blood count normalization), partial response or hematologic improvement (HI). For advanced systemic mastocytosis response is considered a decrease in mast cell burden in bone marrow or serum tryptase level by at least 30%.

# Secondary Objectives:

- To evaluate the safety of GTB-3550 TriKE when administered on this schedule
- To estimate overall survival (OS) at 6 months

# Correlative Objectives:

- To monitor the number, phenotype, activation status and function of NK cells, T cells, T regulatory cells and MDSCs pre- and post-therapy (
- To evaluate the pharmacokinetics and dynamics of the TriKE reagent
- To monitor for the development of human anti-TriKE antibodies
- To monitor the occurrence of antigen negative escape variants ( ) in patients without response

# Eligible Diseases:

Diagnosis of one of the following CD33-expressing myeloid malignancies with greater than or equal to 50% CD33+ target cells with no good standard of care treatment options including:

<u>High Risk Myelodysplastic Syndromes (MDS)</u> progressive on two or more prior regimens and requiring treatment that meets **at least one** of the following:

- IPSS-R High or Very High Risk
- WHO Classification: RAEB-1 or RAEB-2
- Poor and very poor risk cytogenetic abnormality as defined by the IPSS-R cytogenetic classifications
- WHO Based Prognostic Scoring System (WPSS): High or Very High Risk Therapy related MDS and not a candidate for induction chemotherapy or had an inadequate treatment response after induction chemotherapy

Acute Myelogenous Leukemia (AML) meeting at least one of the following:

- Refractory AML defined as failure to achieve remission after at least 3 induction attempts
  - Elderly AML not fit for induction therapy can be enrolled after 2 failed inductions
- Relapsed AML meeting one of the following:
- Not a candidate for hematopoietic stem cell transplant (HSCT), at least one reinduction attempt required
- Prior HSCT relapse beyond 3 months may be included only if off immunosuppression for a minimum of 4 weeks and do not have GVHD

<u>Advanced systemic mastocytosis</u> (defined as mast cell leukemia, aggressive systemic mastocytosis, and systemic mastocytosis associated with hematologic neoplasm) may enroll without any prior treatment, given there is no standard established therapy.

### Key Inclusion Criteria:

- Age ≥ 18 years of age, Karnofsky performance status ≥ 70%
- Adequate renal, hepatic, cardiac and lung function
- Absolute lymphocyte count (ALC) ≥ 200 cells/mm³ OR absolute circulating CD56⁺/CD3⁻ NK cell count >25 cells/µL within the 14 days prior to start of therapy

#### **Enrollment:**

<u>Dose Finding Component:</u> 30 patients enrolled in cohorts of 2 testing up to 7 GTB-3550 TriKE dose levels

#### **Extended Component:**

Stage 1: enroll 13 patients at the MTD (including any from the dose finding component treated at the MTD) – If 3 or more of these 13 patients experience a clinical response by Day 42, the trial will move to Stage 2

Stage 2: enroll 17 additional patients at the MTD established during the dose finding component

If the Phase I component enrolls more than 13 patients at the MTD, the futility rule for the two stage design will be adjusted with the given number of patients enrolled at the MTD.



**Each block consists** of 4 consecutive 24 hour continuous infusion (CI) of GTB-3550 TriKE at the patient's assigned CI dose with a 72 hour rest after Block #1 and #2.

#### **Dose Finding Phase I Component:**

Each patient receives GTB-3550 TriKE at the assigned CI dose for 3 sets (infusion block #1, #2, and #3) of 4 consecutive 24 hours infusions separated by a 72 hour rest.

| Dose<br>Level | GTB-3550 TriKE Dose daily continuous infusion (CI) dose (µg/kg/day) |
|---|---|
| 1 | 5 |
| 2 | 10 |
| 3 | 25 |
| 4 | 50 |
| 5 | 100 |
| 6 | 150 |
| 7 | 200 |

The phase I component uses a continual reassessment method (CRM). Patients are enrolled in cohorts of 2 beginning at Dose Level 1. A minimum of 1 week must separate each patient. Both patients within each cohort must reach Day 28 (end of the DLT assessment period) prior to enrollment of a subsequent cohort. The study statistician assigns each new cohort of 2 patients to the most appropriate dose level based on updated toxicity probabilities. As enrollment proceeds, each cohort will be assigned to an increased, decreased or equivalent dose level based on prior data in the trial. Enrollment continues until the study sample reaches evaluable 30 patients. At that time the maximum tolerated dose (MTD) for the Phase II component will be identified.

**Dose Limiting Toxicity (DLT)** is defined as any related treatment emergent toxicity within 28 days (as assessed on Day 29) of the first dose of TriKE with the exception of those that are clearly and incontrovertibly due to extraneous causes for the following criteria based on CTCAE v5:

- Any Grade 4 or 5 non-hematologic events
- Grade 3 non-hematologic adverse events lasting more than 72 hours, except the following:
  - Non-sustained (< 7 days) Grade 3 liver function tests (ALT/AST, alkaline phosphatase, total or direct bilirubin) abnormalities in the absence of clinical signs of hepatic dysfunction (lethargy, confusion, anorexia, pruritus or tremors).
  - Non-sustained Grade 3 QTc prolongation (< 72 hours) in the absence of cardiac arrhythmia</li>
  - Grade 3 electrolyte disturbances that resolve, with or without intervention, to < Grade 2 levels within 72 hours
  - Grade 3 fatigue
  - o Grade 3 anorexia
  - Grade 3 fever
  - Grade 3 infection

- Hematologic Toxicity Given that AML and MDS inherently leads to low neutrophils and platelets, standard grading cannot be used as many of these patients technically meet criteria for "grade 4" neutropenia or thrombocytopenia at baseline. Thus, the hematologic DLTs are listed below:
  - o AML:
    - Grade 4 neutrophil count (<500/µL) lasting ≥ 29 days from start of cycle in absence of evidence of active leukemia
    - Grade 4 platelet count (<25,000/µL) lasting ≥ 29 days from start of cycle in the absence of active leukemia
    - Any clinically significant bleeding that is not controllable with transfusion support
  - o MDS/mast cell diseases:
    - Grade 4 neutrophil count (<500/µL) lasting ≥ 29 days from start of cycle in absence of evidence of active MDS/mast cell disease
    - Grade 4 platelet count (<25,000/µL) lasting ≥ 29 days from start of cycle in the absence of active MDS/Mast cell disease
    - Any clinically significant bleeding that is not controllable with transfusion support
    - Grade 4 anemia, unexplained by the underlying disease
- Grade 3 infusion related, treatment related reaction including cytokine release syndrome which does not resolve within 72 hours despite best medical management (refer to Section 10 for modified CRS grading)
- Grade 3 or 4 Tumor Lysis Syndrome that does not resolve within 7 days with or without intervention
- Inability to complete at least one block of three 24 hour infusions due to any treatment emergent, treatment related toxicity

**Maximum Tolerated Dose (MTD)** is defined as the dose level that most closely corresponds to the target DLT rate of 20%.

#### Additional Dose Escalation Parameters (Phase I Only):

In addition to monitoring for dose limiting toxicity, patients enrolled in the Phase I component will be monitored for signs of immune activation using treatment related tachycardia and fever as clinical markers of transient bioactivity resulting from endogenous cytokine release. If detected in a single patient, subsequent dose levels will increase by 50% instead of the planned doubling (100% increase).

#### **Extended Phase II Component:**

Patients will receive three consecutive blocks of four 24 hour continuous infusions of GTB-3550 TriKE at the Phase I MTD separated by a 72 hour rest. There is no staggering of enrollment for this component.

**Stage 1**: Enroll a total of 13 patients (including all treated at the MTD in Phase I). If 3 or more of these patients have clinical response by Day 42 the trial will continue to Stage 2. If the Phase I component enrolls more than 13 patients at the MTD, the futility rule for the two-stage design will be adjusted with the given number of patients enrolled at the MTD.

**Stage 2**: Enroll an additional 17 patients. If 10 of 30 patients have a clinical response by Day 42, GTB-3550 TriKE will be considered promising for further investigation.

### Monitoring for Safety (Phase II Extended):

- Grade 4-5 non-hematologic, non-relapse, non-infectious toxicity (except fever) by 42 days after the start of the first GTB-3550 TriKE treatment block
- Non-relapse, non-infectious treatment related mortality within 60 days of the 1<sup>st</sup> dose of GTB-3550 TriKE

# 1 Objectives

### 1.1 Primary Objective

<u>Phase I Dose Finding:</u> To identify the maximum tolerated dose (MTD) of GTB-3550 TriKE defined as the dose level that most closely corresponds to a dose limiting toxicity rate (DLT) of 20%.

<u>Phase II Extension</u>: To determine preliminary efficacy as measured by the rates of "best" clinical response by Day 42 after the start of the 1<sup>st</sup> infusion.

For AML clinical response includes complete remission with or without hematologic or platelet recovery (CR, CRi or CRp) or partial response. For MDS clinical response includes complete remission, marrow CR (with incomplete peripheral blood count normalization), partial response or hematologic improvement (HI). For advanced systemic mastocytosis response is considered a decrease in mast cell burden in bone marrow or serum tryptase level by at least 30%.

## 1.2 Secondary Objectives

- To evaluate the safety of GTB-3550 TriKE when administered on this schedule
- To estimate overall survival (OS) at 6 months

## 1.3 Correlative (Research) Objectives

- To evaluate the phermacolination and dynamics of the Trill research
- To evaluate the pharmacokinetics and dynamics of the TriKE reagent
- To monitor the occurrence of antigen negative escape variants (CD33- blasts) in patients without response

# 2 Background

Acute myeloid leukemia (AML) is a heterogeneous hematologic stem cell malignancy in adults with incidence rate of 3–5% per 100,000 populations. The median age at the time of diagnosis is 65–69 years. AML is an aggressive disease and is fatal without anti-leukemic treatment. Myelodysplastic syndromes (MDS) are a heterogeneous group of myeloid neoplasms characterized by dysplastic features of erythroid/myeloid/megakaryocytic lineages, progressive bone marrow failure, a varying percentage of blast cells, and enhanced risk to evolve into acute myeloid leukemia<sup>3</sup>. The incidence of MDS is rising especially in states like Minnesota for unknown reasons. There are few established treatments for MDS so a drug that could be successfully employed

to treat AML and MDS would be extremely valuable. The expression of cell surface markers in MDS is complicated by its heterogeneous nature and has only been recently brought to light with the work of the First Workshop on Standardization of Flow Cytometry in MDS convened in Amsterdam bringing together experts from Europe, Japan, and the USA<sup>4</sup>. The workshop found that a majority of MDS cases showed an abnormally high expression of HLA-DR, CD64, and CD33. We believe that CD33 is a validated target in AML and can also target MDS cells to promote a novel targeted immunotherapy approach for these diseases.

Targeted cancer immunotherapies are currently a subject of great clinical interest and potential <sup>5</sup>. While a great deal of interest has recently been placed upon generation of chimeric antigen receptor (CAR) expressing T cells from monoclonal antibodies shown to target human malignancies <sup>6</sup>, and more even more recently upon generation of CAR-expressing natural killer (NK) cells <sup>7,8</sup>, these approaches require a personalized approach that is expensive, time consuming, and difficult to apply on a large scale. There is a clear need for targeted off-the-shelf therapies that augment the current monoclonal antibody approach. To accomplish this goal, we focus on generation of tri-specific killer engagers (TriKEs) meant to target NK cells to the tumor synapse and induce their activation at that site. Unlike full-length tri-specific antibodies,



June 4, 2021 



These attributes make them an ideal pharmaceutical platform for potentiated NK cell-based immunotherapies.

# 3 Summary and Rationale

The most important aspects of the humoral (antibody) response against cancer is 1) the ability of antibody to mediated antibody dependent cellular cytotoxicity (ADCC) through CD16, 2) the ability to mediate in vivo expansion of the immune population to recruit more killers to generate an anti-cancer response (the IL-15 linker) and 3) recognition of a target antigen (like CD33 being tested here).

June 4, 2021 



The Trispecific Killer Engager (TriKE) designated GTB-3550 was designed as a straightforward off-the-shelf product that can be used to treat CD33+ AML/MDS patients in a manner similar to the way rituximab is used to treat B cell malignancies. We believe that a major advantage of our drug as compared to chimeric antigen receptor (CAR) transduced T cells that require cell and gene therapy is the simplicity of our approach.

The MTD of exogenous IL-15 in humans following continuous IV infusion is 2 ug/kg/day for a total of 10 days (240 hours).

# 4 Study Design

This is a multisite Phase I/II clinical trial of GTB-3550 (CD16/IL-15/CD33) tri-specific killer cell engager (TriKE) for the treatment of CD33-expressing high risk myelodysplastic syndromes, refractory/relapsed acute myeloid leukemia or advanced systemic mastocytosis. Up to 10 study centers may take part in this trial.

Patients receive a single course of GTB-3550 TriKE given as 3 weekly treatment blocks. Each block consists of four consecutive 24 hour continuous infusions of GTB-3550 TriKE followed by a 72 hour break after Block #1 and #2. All treatment is given as an inpatient.

Toxicities are monitored through Day 28 (as assessed on Day 29) with continued toxicity assessment through Day 60. Disease response is assessed by bone marrow biopsy performed between Day 21 and 42 after the start of the 1st infusion. Follow-up for response and survival continues through 6 months from study treatment start.

The study consists of two components. The dose finding component is a modified version of a Phase I trial and the extended component is a modified Phase II trial.

<u>Dose Finding Component:</u> The Phase I component uses a continual reassessment method (CRM) to determine the maximum tolerated dose (MTD) of GTB-3550 TriKE. Up to 7 doses levels will be tested. The goal of the CRM is to identify the dose level which most closely corresponds to the targeted dose limiting toxicity (DLT) rate of 20%.

Patients are enrolled in cohorts of 2 beginning at Dose Level 1. A minimum of 1 week must separate each patient. Both patients within a cohort must reach Day 28 (end of the DLT assessment period) prior to enrollment of a subsequent cohort. The study statistician assigns each new cohort of 2 patients to the most appropriate dose level based on updated toxicity probabilities. As enrollment proceeds, each cohort is assigned to an increased, decreased or equivalent dose level based on prior data in the trial until the study sample reaches 30. At this time, the last dose is declared the MTD and the GTB-3550 TriKE dose for the extended component.

**Extended Component:** The primary goal of the extended component is to study the potential efficacy of GTB-3550 TriKE in this patient population. Efficacy is measured using rates of complete and partial remission. A Simon's MiniMax two-stage design is used in this phase. Monitoring guidelines are in place to stop the study early for excessive toxicity.

Stage 1 enrolls 13 patients, including all patients treated at the MTD defined during the dose finding component. If 3 or more of these 13 patients have a clinical response to GTB-3550 TriKE, the trial moves to Stage 2 and enrolls an additional 17 patients. If the Phase I component enrolls more than 13 patients at the MTD, the futility rule for the two-stage design will be adjusted with the given number of patients enrolled at the MTD.

If at least 10 of the 30 patients have a clinical response, GTB-3550 TriKE will be considered for further investigation.

Patients experiencing clinical benefit (defined as stable or better) at the time of the 1<sup>st</sup> disease reassessment may be considered for a 2nd course of GTB-3550 TriKE on a compassionate basis provided they experienced no side effects equivalent to a DLT and continue to meet relevant study inclusion/exclusion criteria. Refer to Section 7.4 for additional information.

## 5 Patient Selection

Study entry is open to adult patients 18 years of age and older regardless of gender, race, or ethnic background. While there will be every effort to seek out and include women and minority patients, the patient population is expected to be no different than that of other high risk malignancies studies at the University Of Minnesota and other participating institutions.

A potential participant must meet all of the inclusion and exclusion criteria to be considered eligible for study participation.

# 5.1 Eligible Diseases

Diagnosis of one of the following CD33-expressing myeloid malignancies with greater than or equal to 50% CD33+ target cells with no good standard of care treatment options including:

<u>High Risk Myelodysplastic Syndromes (MDS)</u> progressive on two or more prior regimens and requiring treatment that meets **at least one** of the following:

- IPSS-R High or Very High Risks
- WHO Classification: RAEB-1 or RAEB-2
- Poor and very-poor risk cytogenetic abnormality as defined by the IPSS-R cytogenetic classifications
- WHO Based Prognostic Scoring System (WPSS): High or Very High Risk

<u>Therapy related MDS</u> and not a candidate for induction chemotherapy or had an inadequate treatment response after induction chemotherapy.

Refractory or Relapsed Acute Myelogenous Leukemia (AML) meeting at least one of the following:

- Refractory AML defined as failure to achieve remission after at least 3 induction attempts
  - Elderly AML not fit for induction therapy can be enrolled after 2 failed inductions
- Relapsed AML
  - Not a candidate for hematopoietic stem cell transplant (HSCT), at least one re-induction attempt required
  - Prior HSCT relapse beyond 3 months may be included only if off immunosuppression for a minimum of 4 weeks and do not have GVHD

#### Notes:

- 1) For hypomethylating agents (i.e. decitabine, azacititdine) to count as an induction/re-induction attempt, the patient must have completed a minimum of 3 monthly cycles
- 2) For targeting agents (i.e. sorafenib) to count as an induction/re-induction attempt, the patient must have completed a minimum of 1 month without attaining CR

<u>Advanced systemic mastocytosis</u> (defined as mast cell leukemia, aggressive systemic mastocytosis, and systemic mastocytosis associated with hematologic neoplasm) may enroll without any prior treatment, given there is no standard established therapy.

### 5.2 Age, Performance Status, Organ Function, Contraception Use

- · At least 18 years of age
- Karnofsky score ≥ 70% (Appendix I)
- Adequate organ function within 14 days (30 days for cardiac and pulmonary) of study enrollment defined as:
  - o Renal: an estimated glomerular filtration rate ≥ 60 mL/min/1.73 m<sup>2</sup>
  - Hepatic: AST, ALT, alkaline phosphatase and total bilirubin within normal range
  - Pulmonary function: DLCO corrected (ml/min/mm Hg) defined as no more than 5 units below lower limit of normal (CTCAE v5 Grade 1 carbon monoxide diffusing capacity decreased) based on patient's height, weight, and gender as reported by the institutional pulmonary function lab.
  - o Cardiac: Absence of decompensated congestive heart failure, or uncontrolled arrhythmia; left ventricular ejection fraction ≥ 45% by echocardiogram, MUGA or cardiac MRI.
- Absolute lymphocyte count (ALC) ≥ 200 cells/mm³ OR absolute circulating CD56+/CD3- NK cell count >25 cells/µl within the 14 days prior to start of therapy
- Sexually active females of childbearing potential and males with partners of child-bearing potential must agree to use adequate birth control during study treatment
- Participant provides voluntary written consent signed before performance of any study-related procedure not part of normal medical care

### 5.3 Exclusion Criteria

- New or progressive pulmonary infiltrates on screening chest x-ray or chest CT scan unless cleared for study by Pulmonary. Infiltrates attributed to infection must be stable/improving with associated clinical improvement after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
- Uncontrolled bacterial, fungal or viral infections, known history of HIV
- Active Hepatitis B or Hepatitis C (virus detectable by PCR) chronic asymptomatic viral hepatitis is allowed
- Other concurrent active cancer within the last year (excluding non-melanoma skin cancers)
- Severely clinically obese patients, BMI >38

- Currently taking any over-the-counter [OTC], vitamin, mineral, or dietary supplement within 14 days prior to study drug administration on Day 1 and during study conduct that may confound study safety goals (e.g. St. John's wort). Questions should be discussed with GT Biopharma.
- Pregnant or breast feeding. The effect of GTB-3550 TriKE on the fetus is unknown. Females of childbearing potential must have a blood test within 7 days prior to enrollment to rule out pregnancy - must be repeated if not within 7 days of treatment initiation
- History of central nervous system malignancy or symptoms of active CNS disease
- A family history of long QT syndrome or with a QTc interval > 480 msec at screening
- Currently taking medications known to prolong QT/QTc interval as the potential risk of QT/QTc prolongation is unknown in humans (refer to Appendix V for a list of prohibited medications for eligibility)
- A candidate for potentially curative therapy, including hematopoietic cell transplant
- Unwilling to remain within a 90 minute drive of the study center through at least Day 29

# 6 Patient Screening and Study Enrollment

Written consent must be obtained prior to the performance of any research related tests or procedures. Consent is usually obtained before final eligibility is determined.

# 6.1 Consent and Study Screening in

Any patient who has been consented is to be entered in by the Study Coordinator or designee. If a patient is consented but is not enrolled in the study treatment, the patient's record is updated in as a screen failure and reason for exclusion recorded.

# 6.2 Prior and Concomitant Therapy:

All non-study medications, including prescription, OTC, or herbal therapies, used by the patient will be documented (i) for the 14 days prior to screening (prior medications), (ii) during screening, and (iii) throughout the study (concomitant medications). The Investigator in communication with the Sponsor will review and determine if prior/concomitant medication(s) affect the patient's eligibility to participate or continue to participate in the study.

Administering medications known to elevate Liver Function Tests (LFTs) during the treatment interval and the week before should be avoided. Azole antifungal agents frequently increase liver function tested in >10% of subjects. For 1 week prior to and concurrent with GTB-3550 administration, patients should be treated with micafungin if medically indicated.

## 6.3 Study Enrollment and GTB-3550 TriKE Dose Level

To be eligible for this study, the patient must sign the treatment consent and meet each inclusion criteria and none of the exclusion criteria listed on the eligibility checklist based on the eligibility assessment documented in the patient's medical record.

To complete enrollment in \_\_\_\_\_, the Study Coordinator or designee records the GTB-3550 TriKE dose level assignment.

## 6.4 Inability to Begin Study Treatment

If a patient is enrolled to the study, and is later found not able begin the study treatment, for whatever reason, the patient will be taken off study and treated at the physician's discretion. The Study Coordinator or designee will update of the patient's non-treatment status. The patient will be replaced to fulfill enrollment requirements.

### 6.5 Re-Treatment Enrollment onto 2015LS167R

Any patient, in the judgement of the Principal Investigator, who experiences lack of disease progression or evidence of clinical improvement after completion of the 1st treatment course may be considered for retreatment per Section 7.4. To be eligible for re-treatment the patient must sign the re-treatment consent and meet each inclusion criteria and none of the exclusion criteria listed on the eligibility checklist based on the eligibility assessment documented in the patient's medical record. Any qualifying patient who has signed the re-treatment consent is entered onto the re-treatment protocol ( ) in by the Study Coordinator or designee.

### 7 Treatment Plan

In order to provide optimal patient care and to account for individual medical conditions, investigator discretion may be used in the prescribing of all supportive care drug therapy (i.e. acetaminophen, diphenhydramine, G-CSF, antimicrobials, etc.).

### 7.1 GTB-3550 TriKE Administration

Patients receive a single course of GTB-3550 TriKE at their assigned dose as 3 weekly treatment blocks. Each block consists of four consecutive 24 hour

continuous infusions (over approximately 96 hours) of GTB-3550 TriKE followed by a 72 hour break after Block #1 and #2. All treatment is given as an inpatient.

The assigned dose will be calculated on a weight obtained within 5 days prior to or on day of the 1<sup>st</sup> dose. The dose is not be recalculated for subsequent treatment blocks.

The institutional Investigational Pharmacy will prepare each 24 hour bag for infusion per Section 9.6 based on the patient's assigned GTB-3550 TriKE dose. Each assigned dose will be administered as a 100 mL infusion over 24 hours period at 4.17 mL/hour rate. Note: actual bag volume is 130 ml to allow for the product sample collection before and after infusion.

#### Pre-meds:

Pre-meds: 30 minutes prior to each infusion, patients will receive acetaminophen 325 mg PO and diphenhydramine 25mg PO/IV. Repeat prn.

### IV Fluid Management:

IV fluids should be administered at a minimum rate of 50 cc/hour additional fluids given based on the clinical status of the patient.

### **Infusion Related Reactions:**

If Grade 2 infusion related reaction occurs, interrupt the infusion and treat symptomatically with antihistamines, NSAIDS, narcotics, IV fluids as medically appropriate. Any patient experiencing a second Grade 2 infusion related reaction after restarting, despite pre-medication or a Grade 3 or 4 infusion related reaction will be permanently discontinued from GTB-3550 TriKE.

Administration of glucocorticoids is prohibited during the TriKE treatment period as the use of systemic steroid medications may result in loss of therapeutic effects of the study drug. They should be avoided except in the event of a severe toxicity.

Any Grade 3 or 4 infusion related reaction will result in permanent discontinuation of study drug with appropriate medical intervention.

### Post-Infusion TriKE Sample Collection (Week 1 infusions only):

Upon completion of <u>each</u> infusion during Week 1 only, the nursing staff will disconnect the infusion bag and tubing from the patient. Prior to discarding the bag and tubing, two pre-labeled 1.8 ml cryo-vial (containing wording "Post-Infusion" as well as dose and date when bag was prepared) will be filled with a minimum of 1 ml of drug each. This may be done on the unit or the bag/tubing transferred to the institutional research lab and samples collected there. Regardless, the vials or

infusion bag/tubing must be refrigerated while awaiting transfer to the research lab. The research lab will freeze samples for later batch shipping to UMN TTL (if applicable) and testing. Refer to Section 8.2 for additional details.

June 4, 2021 

## 7.1.1 Monitoring Requirements During TriKE Infusions

## Monitoring during the 1<sup>st</sup> infusion of each continuous infusion (CI) block:

Vital signs including blood pressure, pulse, temperature, respirations, and pulse oximetry will be measured as follows:

- prior to the infusion start
- every 15 minutes (±10 minutes) during the 1<sup>st</sup> hour
- every 30 minutes (±10 minutes) during the 2<sup>nd</sup> hour
- every 60 minutes (±10 minutes) for the next 2 hours
- then every 4 hours (±20 minutes) for the remainder of the infusion

### Monitoring during the infusion 2, 3, and 4 of each CI block:

Vital signs including blood pressure, pulse, temperature, respirations, and pulse oximetry will be measured as follows:

- every 15 minutes (±10 minutes) during the 1<sup>st</sup> hour
- then every 4 hours (±20 minutes) for the remainder of the infusion

Targeted toxicities (Appendix VI) and unexpected adverse events will be collected at the time points listed in Section 10.2.

### 7.1.2 Monitoring for Signs of Immune Activation (Phase I Patients):

In addition to monitoring as above, patients enrolled in Phase I will be monitored for clinical signs of immune activation:

- treatment related tachycardia defined as a heart rate of >30 BPM than baseline heart rate measured each cycle pre-infusion and persists for 4 hours
- fever defined as Grade 2 (>39.0 40.0 degrees C [102.3 104.0 degrees
   F]) and persists for 4 hours

If a patient meets either of the above criteria, no dose adjustment will be made unless a dose limiting toxicity (DLT) occurs. Refer to Section 7.2.1 for impact on subsequent dose level escalation.

### 7.1.3 Supportive Care/Concomitant Medications

Supportive measures may include acetaminophen for fevers, meperidine for chills, anti-emetics for nausea and vomiting, normal saline or furosemide to maintain fluid balance/blood pressure/pulmonary function, and electrolyte replacement. Use of G-CSF is permitted as clinically indicated. Refer to Section 7.3 for management of selected toxicities.

Administration of glucocorticoids is prohibited during the TriKE treatment period as the use of systemic steroid medications may result in loss of therapeutic effects of the study drug. They should be avoided except in the event of a severe toxicity.

The potential risk of QT/QTc prolongation is unknown in humans receiving TriKE. Persons with a family history of long QT syndrome, with a QTc interval > 480 msec at screening, or taking concurrent medications known to prolong QT/QTc interval are not eligible for this study. The use of medications known to prolong QT/QTc interval (refer to Appendix V) are prohibited between screening and the end of treatment visit if at all possible.

The interactions between TriKE and the P450 system are unknown. The IL-15 component may affect substrates of CYP3A4 and CYP2D6 substrates. See Appendix IV for a list of drugs which may be affected. Patients with unexpected toxicity should have a review of their con-meds to determine whether there are any potential interactions. The PI or treating physician should consider discontinuing these medications as clinically indicated.

All concomitant medications, with a start and stop date must be documented relative to administration of GTB-3550 TriKE.

### 7.1.4 Dose Modifications

No individual patient dose modifications are permitted other than as described in Section 7.3.3 for elevated liver enzymes.

### 7.1.5 Criteria to Continue with GTB-3550 TriKE Block #2 and #3

A dose limiting toxicity (for any patient, not just dose finding) during the previous block's infusions (defined in Section 7.2.1) will disqualify a patient from receiving further therapy.

**Disease based treatment decisions:** If after completing Block #1 and Block #2, the patient has clear evidence of disease progression they will be discontinued from study treatment and further treatment with study drug is to be discontinued. Such patients remain fully evaluable for efficacy and toxicity.

To begin a new block, on the day of the planned treatment the patient must:

- not currently meet any disease specific hematologic dose limiting toxicity as defined in Section 7.2.1.
- have an estimated glomerular filtration rate ≥ 60 mL/min/1.73 m<sup>2</sup>
- have a total bilirubin of ≤1.5 times the ULN

- have AST and ALT ≤ 3 x upper limit of normal, and alkaline phosphatase levels ≤ 2.5 x upper limit of normal
- be afebrile (defined as a temperature of ≤ 101°F)
- have room air 0₂ saturation ≥ 88%
- have a blood pressure ≥ 100/65 mm/Hg
- have no signs or symptoms of infection

If the above criteria is not met, treatment must be delayed for appropriate supportive care and clinical assessment. The study drug may begin the following day, if the above criteria are met and, in the opinion of the clinical provider it is safe to proceed. Otherwise delay 1 week from the planned start and reassess at that time.

Patients unable to begin treatment after a 1 week delay will be permanently discontinued from treatment and followed per Section 7.6.

The start of Block #2 or Block #3 may be delayed for up to 1 week (i.e. start 1 week later than planned) to allow for the resolution of any treatment or non-treatment issues (i.e. URI, UTI, etc.) or for holiday/scheduling issues.

### 7.2 GTB-3550 TriKE Dose Levels

### 7.2.1 Dose Finding Component (Phase I)

The 1<sup>st</sup> two patients will be assigned dose level 1. The study statistician (UMN biostatistician Todd DeFor or designee) will assign each new cohort of 2 patients to the most appropriate dose level based on updated toxicity probabilities. Both patients within a dose cohort must reach Day 28 (end of the DLT assessment period) prior to enrollment of a subsequent cohort. Enrollment continues until 30 evaluable patients are accrued.

| Dose<br>Level | GTB-3550 TriKE Dose<br>daily continuous infusion<br>(CI) dose (µg/kg/day) |
|---|---|
| 1 | 5 |
| 2 | 10 |
| 3 | 25 |
| 4 | 50 |
| 5 | 100 |
| 6 | 150 |
| 7 | 200 |

**Dose Limiting Toxicity (DLT)** is defined as any of the following related treatment emergent toxicity with the exception of those that are clearly and incontrovertibly due to extraneous causes within 28 days (**as assessed on Day 29**) of the first dose of TriKE for the following criteria based on CTCAE v5:

- Any Grade 4 or 5 non-hematologic events
- Grade 3 non-hematologic adverse events lasting more than 72 hours, except the following:
  - Non-sustained (< 7 days) Grade 3 liver function tests (ALT/AST, alkaline phosphatase, total or direct bilirubin) abnormalities in the absence of clinical signs of hepatic dysfunction (lethargy, confusion, anorexia, pruritus or tremors).
  - Non-sustained Grade 3 QTc prolongation (< 72 hours) in the absence of cardiac arrhythmia
  - Grade 3 electrolyte disturbances that resolve, with or without intervention, to < Grade 2 levels within 72 hours</li>
  - o Grade 3 fatigue
  - Grade 3 anorexia
  - Grade 3 fever
  - Grade 3 infection
- Hematologic Toxicity Given that AML and MDS inherently leads to low neutrophils and platelets, standard grading cannot be used as many of these patients technically meet criteria for "Grade 4" neutropenia or thrombocytopenia at baseline. Thus, the hematologic DLTs are listed below:
  - o AML
  - Grade 4 neutrophil count (< 500/µL) lasting ≥ 29 days from start of cycle in absence of evidence of active leukemia
  - Grade 4 platelet count (< 25,000/uL) lasting ≥ 29 days from start of cycle in absence of evidence of active leukemia

Any clinically significant bleeding that is not controllable with transfusion support

- MDS/mast cell diseases:
- Grade 4 neutrophil count (<500/µL) lasting ≥ 29 days from start of cycle in absence of evidence of active MDS/mast cell disease
- Grade 4 platelet count (<25,000/µL) lasting ≥ 29 days from start of cycle in the absence of active MDS/Mast cell disease
- Any clinically significant bleeding that is not controllable with transfusion support
- Grade 4 anemia, unexplained by the underlying disease

- Grade 3 infusion related, treatment related reaction including cytokine release syndrome which does not resolve within 72 hours despite best medical management (refer to Section 10 for modified CRS grading)
- Grade 3 or 4 Tumor Lysis Syndrome that does not resolve within 7 days with or without intervention
- Inability to complete at least one block of three 24 hour infusions due to any treatment emergent, treatment related toxicity.

**Maximum Tolerated Dose (MTD)** is defined as the dose level that most closely corresponds to the target DLT rate of 20%.

### Additional Dose Escalation Parameters (Phase I Only):

In addition to monitoring for dose limiting toxicity, patients enrolled in the Phase I component will be monitored for signs of immune activation using treatment related tachycardia and fever as clinical markers of transient bioactivity. Refer to Section 7.1.2 Monitoring for Signs of Immune Activation (Phase I patients) for the definition of tachycardia and fever thresholds.

If detected in a single patient (fever or tachycardia lasting > 4 hours OR meets criteria for any DLT) subsequent dose levels will increase by 50% instead of the planned doubling (100% increase). For example, if signs of immune activation occurred at Dose Level 4 (50  $\mu$ g/kg/day), Dose Level 5 would be adjusted to 75  $\mu$ g/kg/day rather than 100  $\mu$ g/kg/day and Dose Level 6 would be 115  $\mu$ g/kg/day (75 x 1.5 rounded up to the nearest 5) rather than 200  $\mu$ g/kg/day.

### 7.2.2 Extended Component (Phase II)

The treatment schedule is identical to the dose finding component. The extended component uses a Simon's MiniMax two-stage design for continued enrollment using the maximum tolerated dose (MTD) established during Phase I with monitoring guidelines to stop the study early for excessive toxicity.

In Stage 1, a total of 13 patients (including all treated at the MTD in part 1) will be enrolled. If 3 or more of these have clinical response the trial will continue to Stage 2. If the phase I component enrolls more than 13 patients at the MTD, the two-stage design will be adjusted with the given number of patients enrolled at the MTD.

In Stage 2, an additional 17 patients will be enrolled for a total of 30 patients treated at the MTD.

### 7.3 Management of Selected GTB-3550 TriKE Toxicities

Throughout the study, the investigator may prescribe any concomitant medications or treatment deemed necessary to provide adequate supportive care. Supportive care may include antibiotics, anti-fungals, analgesics, transfusions, and G-CSF/cytokines.

Note: Any patient experiencing a DLT equivalent toxicity must discontinue treatment per Section 7.5 and is not eligible for retreatment.

Please refer to Section 9.7 for potential toxicities.

### 7.3.1 Tumor Lysis Syndrome

Tumor lysis syndrome is a possible risk associated with therapy of active leukemia. All patients (except those with known allergy) will begin on prophylactic allopurinol 300 mg po before the 1<sup>st</sup> dose of GTB-3550 TriKE and continue daily as clinically indicated.

### 7.3.2 Infusion Related Reaction

Patients will be monitored for the occurrence of hypotension, dyspnea and angioedema during the infusion. The infusion will be stopped and the reaction treated per Section 7.1. A Grade 3 or Grade 4 infusion related reaction will result in permanent discontinuation of the infusion.

#### 7.3.3 Increase in Liver Function Tests

Liver function tests will be monitored three times weekly during each CI block and at Day 22, 29, and 60 visits.

Elevated liver function tests (ALT, AST and/or total bilirubin) guidelines based on CTCAE v 5 grading:

### **Grade 1 or 2:** continue therapy per protocol

**Grade 3:** discontinue treatment for the current block after completion of the currently hung infusion bag, if applicable. Missed doses are not made up.

At the time of next scheduled treatment, if LFTs return to Grade 0 in two weeks or less, initiate the next block of treatment; however, reduce the TriKE dosing by 1 dose level.

**Grade 4 or recurrence of a Grade 3**: permanently discontinue therapy

### 7.3.4 Neurotoxicity

A neurological assessment including basic motor (gait), coordination (steadiness) and cognitive function (alert and oriented) should be performed daily during each CI block. Any abnormalities should be followed up with a detailed neurologic exam and appropriate clinical care.

### 7.3.5 Pulmonary Toxicity

Patients will be monitored for clinical signs and symptoms of pulmonary toxicity through routine daily patient assessments and via the Targeted Toxicities Worksheet (Appendix VI). O<sub>2</sub> saturation levels will be checked per routine in-patient assessments (minimum of once every nursing shift).

Any new hypoxia will be evaluated with a chest x-ray or other imaging as clinically indicated.

Grade 3 hypoxia (decreased oxygen saturation at rest [e.g., pulse oximeter < 88%]) or higher is a dose limiting toxicity. In this situation, discontinue treatment for per Section 7.5 after completion of the currently hung infusion bag, if applicable.

### 7.3.6 Cytokine Release Syndrome (CRS) or CRS-Like Symptoms

While CRS is a clearly defined syndrome in T cell therapy, it is not known to occur to the full extent in NK cell therapies. However, we have seen immune activation syndromes with other IL-15 products that include fever, and rash. If symptoms occur, CRP, IL-6 and ferritin levels will be assessed. If indicated by the presence of medically significant symptoms and/or high IL-6 levels or any symptoms requiring intervention, steroids are the first line of treatment.

Patients will be monitored for clinical signs and symptoms of CRS through routine daily patient assessments and via the Targeted Toxicities Worksheet (Appendix VI). Refer to Section 10 for the revised CRS grading system that will be used for this study.

# 7.4 Opportunity for Re-Treatment

If a patient completes the planned 3 blocks of TriKEs treatment per protocol with lack of disease progression or evidence of a clinical improvement, re-treatment may be an option after discussion with the institutional PI or designee. The patient must continue to fulfill the relevant eligibility criteria in Section 5 and have had no toxicity equivalent to a DLT with the 1st treatment course. Participants would sign a re-treatment consent and be enrolled onto the retreatment protocol CPRC
#2015LS167R, while continuing to be followed for the main study's endpoints as planned.

Eligible patients will receive TriKE at the same or a lower dose level and on the same schedule as initially treated. Treatment must begin within 2 to 4 weeks after completion of the 1<sup>st</sup> course. Treatment guidelines will be followed per Section 7. Re-treatment patient events will not apply toward dose limiting toxicities (DLTs) or early stopping rule events. Tests and evaluations (with a limited research related sample collection plan) during and after treatment would follow those in Section 8.1 and Section 8.3. This includes frequent assessments for toxicity and survival follow-up through 6 months from the 1<sup>st</sup> dose of the re-treatment.

Such situations are considered compassionate and would not be included in the statistical analysis.

### 7.5 Duration of Study Treatment

Patients will receive one treatment course consisting of three sets (blocks) of four consecutive 24 hour continuous infusions GTB-3550 TriKE unless:

- the patient experiences the equivalent of a dose limiting toxicity (see Section 7.2.1 for definition),
- the patient is unable to start Block #2 or #3 within 1 week of the planned date.
- the patient refuses further treatment,
- Disease based treatment decisions: If after completing Block #1 and Block #2, the patient has clear evidence of disease progression they will be discontinued from study treatment and further treatment with study drug is to be discontinued.
- In the opinion of the treating investigator, continuing treatment is not in the best interest of the patient.

For patients discontinuing prior to completing 3 blocks, post-treatment activities at Day 22 and Day 29 are shifted earlier to maintain the timing (i.e. 1 and 2 weeks from the start of the final block).

### 7.6 Duration of Study Participation

Direct study participation ends with the end of treatment visit at Day +60 (±1 week) or earlier, if a new treatment is started. For patients not receiving all 3 blocks, the end of treatment visit occurs approximately 6 weeks (±1 week) from the start of the last block.

Further treatment, independent of the study, will be at the treating physician's discretion.

Follow-up will continue for overall survival continues on all evaluable patients through 6 months from the 1<sup>st</sup> treatment by record review or other means.

### 8 Schedule of Patient Activities

Scheduled evaluations after screening may be performed ±1 day from the targeted date through Day 29; unless otherwise noted. A disease reassessment will occur between Days 21 and 42. A ±7 day window is permitted for the end of treatment (EOT) visit. If a patient discontinues treatment before receiving all 3 blocks, subsequent time points are adjusted to maintain timing (i.e. Day 22 is moved to 1 week after the start of the last block).

In addition, targeted days may be altered as clinically appropriate. Follow-up visits are per standard of care with disease status and survival status abstracted from the medical record.

### 8.1 Required Standard of Care

Standard of care procedures should be followed for all enrolled patients, including those who are enrolled for retreatment.

| Activity | Screening within 30 days of enrollment (within 14 days if for eligibility) | Day 1, Day 8, and Day 15 (start of treatment block) | Daily<br>during<br>infusions<br>(i.e. Day 2-5,<br>9 12, 16-19) | Day<br>22 | Day<br>29 | Anytime<br>between<br>Day 21<br>through<br>Day 42 | End of<br>Treatment<br>Visit<br>Day 60<br>(±7 days) | FU for<br>overall<br>survival<br>(through<br>Month 6) |
|---|---|---|---|---|---|---|---|---|
| consent | X | ысыку | 0 12, 10 10) | | | Day IL | (±1 days) | Wioriti 0) |
| baseline | X | | | | | | | |
| assessment | ^ | | | | | | | |
| medical history | Х | X | | | Х | | Х | |
| concomitant meds <sup>7</sup> | X | X | Х | X | X | | X | |
| concomitant meds | | | Χ | | | | | |
| physical exam | X | X | | Χ | Χ | | X | |
| vital signs including pulse oximetry | Х | Х | per<br>Section 7.1.1 | Х | Х | | Х | |
| neurologic | | _ | X | | | | | |
| assessment | | $X^2$ | ^ | | | | | |
| provider assessment | | | X | | - | | | |
| | | | ^ | | | | X <sup>5</sup> | ~ |
| survival status | | X | X | | - V | | | X |
| assessment of toxicity | | X | Χ | Х | X | | X | |
| Karnofsky PS | X | | | | Х | | Х | |
| height | X | | | | | | | |
| weight | | X (- 5 days) | | | | | | |
| CBC/diff/plt | X | X | X | X | Х | | Х | |
| basic metabolic | | | X | | | | | |
| panel | | | | | | | | |
| comprehensive | | | | | | | | |
| metabolic panel <sup>3</sup> , | X | X | | Х | Х | | X | |
| magnesium and | | χ | | ^ | | | | |
| phosphorus | | | | | | | | |
| ALT, AST, total bili, | | | 2 times | | | | | |
| albumin <sup>4</sup> | | | Z times | | | | | |
| hepatitis B and C | × | | | | | | | |
| screening | ^ | | | | | | | |
| INR <sup>8</sup> | Х | | | | | | | |
| eGFR | Х | | | | | | | |
| Serum pregnancy test | | | | | | | | |
| for FOCBP within 7 | X | | | | | | | |
| days of treatment star | | | | | | | | |
| Disease assessment | Х | | | | | Х | | |
| BM biopsy <sup>1</sup> | X | | | | | X | | |
| Electrocardiogram | X | | | | | | | |
| Echocardiogram, | X | | | | | | | |
| cardiac MRI or | | | | | | | | |
| MUGA | | | | | | | | |
| Chest/abdomen CT | Х | | | | | | | |
| assessment of | | | | | 1 | | | |
| response | | | | | | Х | | $X^6$ |
| 1 - sample to TTI per S | Cootion 0.2 of tin | as of each SOC | hana marrau h | ionov | 1 | I | 1 | 1 |

<sup>1 -</sup> sample to TTL per Section 8.2 at time of each SOC bone marrow biopsy

June 4, 2021 

<sup>2 -</sup> Neurological assessment daily including basic motor (gait), coordination (steadiness) and cognitive function (alert and oriented) - any abnormalities should be followed up with a detailed neurologic exam.

<sup>3 -</sup> Albumin, alkaline phosphatase, ALT, AST, bilirubin (total), calcium, chloride, CO2, creatinine, glucose, potassium, protein (total), sodium, urea nitrogen

<sup>4 -</sup> perform LFTs and albumin twice more during infusion week (in addition to Day of infusion start CMP) = three times during infusion week

- 5 survival status at Day 60 for early study stopping rule for expansion component only
- 6 until relapse/progression or start of a new therapy, then survival only
- 7 document all concomitant medications, including start and stop dates, relative to administration of GTB-3550 TriKE
- 8- Measure and report prior to commencement of GTB-3550 therapy for information only and not as criteria for inclusion.

June 4, 2021 

### 8.2 Research Related Testing, Assessments, and Sample Collections

Sample collections and other procedures after the end of the infusions will coincide with outpatient clinic visits which may not occur on the targeted day.

| | Screen/ | Pre Dose 1<br>each Block | Daily during infusions (i.e. Day 2-5, 9-12, 16- | | | Day | Day of SOC Disease Reassessmen t (Day 21 – |
|---|---|---|---|---|---|---|---|
| | Baseline | (Day 1, 8, 15) | 19) | block | 22 | 29 | Day 42) |
| Toxicity Assessment | | (= =-) -, -, -,, | , | ction 10.2 for det | | | |
| Assessment for dose | | Bv Dav 29 - | report as DLT for Phase | | | ent | |
| limiting toxicity | | | DLT is not eligible to cont | | | | |
| Assessment for | | Expansion co | omponent only through D | ay 42 for non-he | ematolog | gic, non- | relapse, non- |
| stopping rules | | | infectious toxicity (ex | cept fever), Day | 60 for T | RM, | |
| Monitoring for signs of | | Pre and during | g TriKE infusions – all | | | | |
| immune activation | | 1 | patients | | | | |
| CRP, ferritin <sup>4</sup> | X | Х | X (Day 5 only) | | | | |
| Pulmonary Function<br>Testing | Х | | | | | | |
| EKG | | X<br>(At 4 hours<br>(±15 min) into<br>the infusion) | X (at 4 hours (±15 min) into each daily infusion and at 4 hours (±15 min) after disconnect at block end) | | | | |
| T Cell Subset | Х | | | | | | |
| Extended Profile <sup>4</sup> | ^ | | | | | | |
| 5 - 10 ml green top | | | X | | | | |
| tubes and 1- 10 ml red top tube | Χ | X | (Day 3, 10, and 17,<br>only)⁵ | | Х | Х | X <sup>3</sup> |
| antibody testing (sample obtained from the 10 ml red top collected in previous row) | <b>X</b> <sup>2</sup> | X (Day 15<br>only) | | | X | x | X <sup>3</sup> |
| 5 ml red top for each PK/PD time point | | Х | х | X¹ | | | |
| 30 ml or as much as able<br>to obtain of heparinized<br>bone marrow aspirate at<br>time of SOC bm bx | X <sup>3</sup> | | | | | | X <sub>6</sub> |
| Pre- and Post-TriKE dru | g product c | oncentrations lev | vels samples – each dru | ug bag during V | Veek 1 | only | |
| TriKE pre-infusion | | | during Week 1 only per | | | | |
| sample - 2 ml of drug | | | - collected after drug | | | | |
| split between two pre- | | preparation is complete and before bag | | | | | |
| labeled 1.8 ml cryo-vials | | sent to floor, – keep refrigerated until pick-up | | | | | |
| TriKE post-infusion | | Each drug bag during Week 1 only – per | | | | | |
| sample collection ~2 ml | | Section 7.1 after infusion end and prior to | | | | | |
| of drug split between two | | discarding ba | | | | | |
| pre-labeled 1.8 ml cryo-<br>vials | | | il samples are collected | | | | |

<sup>1.</sup> PK/PD time points in association with the end of each infusion block (i.e. Day 5, 12, and 19 or at the discontinuation of the block's infusions, if prior to 96 hours) - 1 hour post (±5 min), 2 hours post (±10 min), 3 hours post (±10 min) and optional 10 hours (±30 min)

<sup>2.</sup> Antibody testing will not be performed in real time nor affect a patient's initial eligibility or ongoing treatment

<sup>3.</sup> Baseline sample if feasible (repeat marrow is not required solely for research sample)

- 4. To Institution's clinical lab, charge to research
- 5. A +2 day window is permitted for this time point (Day 3 (window of days 3- 5), Day 10 (window of days 10-12) and Day 17 (window of days 17-19)
- 6. At time of post-treatment bone marrow biopsy or at Day 60 (End of Treatment visit)

**For UMN patients**: All samples unless otherwise noted go to Masonic Cancer Center Translational Therapy Laboratory (TTL) - Call for sample pick-up.

### For non-University of Minnesota sites:

- The 5 green top and 1 red top samples are shipped the day of collection (Monday-Thursday) for next day delivery to the Masonic Cancer Center's Translational Therapy Lab (MCC TTL).
- PK/PD samples are stored frozen and batched shipped to MCC TTL at the end of the patient's treatment.
- TriKE pre and post infusion samples (Week 1 only) are stored frozen and batch shipped to MCC TTL during Week 2.
- Bone marrow aspirate is collected at the time of standard of care bone marrow prior to treatment start and at the time of the post-treatment bone marrow biopsy. Ship day of collection to MCC TTL.

Refer to the Laboratory Manual for additional details.

It is recognized that with novel therapies as used in this study, the timing of protocol directed research samples may miss important patient specific events. For this reason, additional sets of research samples may be drawn at up to 3 time points that are not specified above.

Note: if a patient is not abiding by the standard of care study calendar (Section 8.1), collection of the research related samples (and targeted toxicities) may be altered or discontinued on an individual patient basis, as appropriate.

## 8.3 Re-Treatment Research Related Testing, Assessments, and Sample Collections

All standard of care procedures described in Section 8.1 are also required for retreatment. Sample collections and other procedures after the end of the infusions will coincide with outpatient clinic visits (and may not occur on the targeted day).

| Screen/ Baseline Pre Dose 1 Day 5 TriKE infusions the last of (Day 21 – Day 42) Toxicity Assessment Monitoring for signs of immune activation CRP, ferritin¹ X X X X Pulmonary Function Testing T Cell Subset Extended Profile¹ 5 - 10 ml green top tube and 1- 10 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at time of SOC bm bx Toxicity Refer to Section 10.2 for details Pre and during TriKE infusions – all patients A X X X X X X X X X X X X X X X X X X | | | Block | 1 only | | | Day of SOC |
|---|---|---|---|---|---|---|---|
| Screen/ Baseline Pre Dose 1 Day 5 Pre and during the start of the last block 42) | | | | | | Day 22 or 1 | Disease |
| Toxicity Assessment Monitoring for signs of immune activation CRP, ferritin¹ X X X X Pulmonary Function Testing T Cell Subset Extended Profile¹ X S - 10 ml green top tubes and 1- 10 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at Nefer to Section 10.2 for details Refer to Section 10.2 for details Refer to Section 10.2 for details Refer to Section 10.2 for details At 2 Refer to Section 10.2 for details At 3 A X X X X X X X X X X X X X X X X X X | | , | | | | | |
| Toxicity Assessment Monitoring for signs of immune activation CRP, ferritin¹ X X X X Pulmonary Function Testing T Cell Subset Extended Profile¹ X 5 - 10 ml green top tube antibody testing 5 ml red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | | - | | 5 - | • | | ` ' |
| Assessment Monitoring for signs of immune activation CRP, ferritin¹ X X X X Pulmonary Function Testing T Cell Subset Extended Profile¹ X 5 - 10 ml green top tube and 1- 10 ml red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | | Baseline | Pre Dose 1 | Day 5 | Trike infusions | the last block | 42) |
| Monitoring for signs of immune activation CRP, ferritin¹ X X X X Pulmonary Function Testing T Cell Subset Extended Profile¹ X 5 - 10 ml green top tubes and 1- 10 ml red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | • | | | | Refer | to Section 10.2 f | or details |
| of immune activation CRP, ferritin¹ X X X X X | | | | | | | |
| activation CRP, ferritin¹ X X X X Pulmonary Function Testing T Cell Subset Extended Profile¹ X 5 - 10 ml green top tubes and 1- 10 ml red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | | | | | | | |
| CRP, ferritin¹ X X X X X Pulmonary Function Testing X T Cell Subset Extended Profile¹ X X X X X X X X X X X X X X X X X X X | | | | | Pre and duri | ng TriKE infusio | ns – all patients |
| Pulmonary Function Testing T Cell Subset Extended Profile¹ 5 - 10 ml green top tubes and 1- 10 ml red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | | | | | | | |
| Function Testing T Cell Subset Extended Profile¹ 5 - 10 ml green top tubes and 1- 10 ml red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | CRP, ferritin <sup>1</sup> | Х | X | X | | | |
| T Cell Subset Extended Profile¹ 5 - 10 ml green top tubes and 1- 10 ml red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | Pulmonary | V | | | | | |
| Extended Profile¹ 5 - 10 ml green top tubes and 1- 10 ml | Function Testing | ^ | | | | | |
| Extended Profile¹ 5 - 10 ml green top tubes and 1- 10 ml red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | T Cell Subset | V | | | | | |
| tubes and 1- 10 ml red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | Extended Profile <sup>1</sup> | ^ | | | | | |
| red top tube antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | 5 - 10 ml green top | | | | | | |
| antibody testing 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | tubes and 1- 10 ml | | X | | | X | |
| 5 ml red top tube (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | red top tube | | | | | | |
| (sample obtained from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | antibody testing | | | | | | |
| from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at | 5 ml red top tube | | | | | | |
| from the 10 ml red top collected in previous row) 30 ml or as much as able to obtain of heparinized bone X3 X marrow aspirate at | (sample obtained | V2 | | | | V | |
| previous row) 30 ml or as much as able to obtain of heparinized bone marrow aspirate at X X | from the 10 ml red | X- | | | | Χ | |
| 30 ml or as much as able to obtain of heparinized bone marrow aspirate at X X | top collected in | | | | | | |
| as able to obtain of heparinized bone X3 X X | previous row) | | | | | | |
| heparinized bone marrow aspirate at X3 X | 30 ml or as much | | | | | | |
| heparinized bone X marrow aspirate at X | as able to obtain of | <b>v</b> 3 | | | | | |
| | heparinized bone | ^~ | | | | | X |
| time of SOC bm bx | marrow aspirate at | | | | | | |
| | time of SOC bm bx | | | | | | |

<sup>1-</sup> To Institutional Lab, but charge to research

For UMN patients, all samples unless otherwise noted go to Masonic Cancer Center Translational Therapy Laboratory (TTL) - Call for sample pick-up.

For non-University of Minnesota sites, refer to Section 8.2 for shipping information.

All "rules" of sample collection found in Section 8.2 also apply to the re-treatment research samples (i.e., windows, missed samples, extra samples).

June 4, 2021 

<sup>2-</sup> Antibody testing will not be performed in real time nor affect a patient's initial eligibility or ongoing treatment

<sup>3-</sup> May be same sample as reassessment from 1st treatment course

### 8.4 Overview of Planned Correlative Studies

A number of correlative studies are performed to understand the safety and ability of the GTB-3550 TriKE to activate the immune response. Immune monitoring is a critical component of the GTB-3550 TriKE clinical trial to understand the drug pharmacokinetic/pharmacodynamic (PK/PD), its in vivo functional activity and clinical tolerance.

- 1. PK sampling to determine TriKE levels and secondary cytokines. In association with each TriKE treatment block, TriKE concentrations will be determined at multiple time points by standard IL-15 ELISA to detect the IL-15 linker in the TriKE as we have already validated. Samples will also be contract tested for IFNα, IL-6, IL-10 and TNF (and other inflammatory cytokines determined informative). This will allow us to determine drug PK/PD and immediate secondary cytokine responses in vivo.
- 2. Determine the absolute number and proportion of NK cells, T cells and their subsets. We have designed multi-color flow cytometry panels to look at basic lymphocytes in whole blood as well as in more detail on ficolled mononuclear cells to determine lymphocyte (and subset) proliferation as measured by Ki-67, inhibitory cells [Treg and CD33+ myeloid-derived suppressor cells] and a number of established NK cell subsets defining adaptive or conventional NK cells.
- NK cell function induced by GTB-3550 TriKE. CD107A degranulation and cytokine production against K562 (to measure natural cytotoxicity) and CD33+ HL60 targets (± exogenous TriKE) will be performed.



5. Pre- and Post- TriKE drug product concentrations levels samples will be stored in TTL frozen at < -70°C for future batch testing.

The marrow will be used in the research lab to study CD33 expression and targeting by allogeneic and autologous lymphocytes.

### 9 GTB-3550 TriKE Description, Supply, Preparation, and Potential **Toxicities**



June 4, 2021 

# 9.5 Study Site Storage and Product Stability 9.6 Preparation and Administration

June 4, 2021 



### 9.7 Potential Toxicities

Although blinatumomab, a bi-specific T cell engager (BiTE), is conceptually similar to our NK cell GTB-3550 TriKE, there are important differences. Blinatumomab's toxicity is presumed related to the anti-CD3 moiety that acts as a potent stimulus for CD3+ T cells. The TriKE is different since the anti-CD16 moiety does not deliver a proliferative stimulus and in fact, we do not expect that promotion of an immune synapse alone will lead to toxicity much like natural engagement of CD16 by FDA-approved monoclonal antibodies such as trastuzumab or rituximab. Instead, we expect the toxicities of GTB-3550 TriKE may be similar to those seen with blinatumomab and/or IL-15. Other than the intramural center at the NCI in Washington DC, we probably have the most experience administering IL-15 to patients as a single agent and in combination with chemotherapy and NK cells.

Most of the side effects of IL-15 are related to immune activation including fevers, chills and some degree of immune activation. We have a prospective plan to monitor patients for these immune side effects to characterize the safety profile of the TriKE. In addition, we will use fever and tachycardia as validated clinical markers to measure early signs of immune activation to modify our dose escalation plan if needed.

June 4, 2021 

### 10 Event Monitoring, Documentation and Reporting

Toxicity and adverse events will be classified according to NCI's Common Terminology Criteria for Adverse Events version 5 (CTCAE v5). A copy of the CTCAE can be downloaded from the CTEP home page at

https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/CTCAE\_v 5\_Quick\_Reference\_5x7.pdf

An exception to the use of CTCAE will be for the assessment of cytokine release syndrome (CRS). Individual adverse events which are associated with CRS will be graded per CTCAE; however the ultimate assessment will be made using a revised grading system for CRS as presented by Lee et al<sup>43</sup>.

| | CRS Revised Grading System (replaces CTCAE v4 CRS grading) |
|---|---|
| Grade | Toxicity Description |
| Grade 1 | Symptoms are not life threatening and require symptomatic treatment only, e.g., fever, nausea, |
| | fatigue, headache, myalgias, malaise |
| Grade 2 | Symptoms require and respond to moderate intervention - Oxygen requirement < 40% or |
| | Hypotension responsive to fluids or low dose of one vasopressor or Grade 2 organ toxicity |
| Grade 3 | Grade 3 Symptoms require and respond to aggressive intervention - Oxygen requirement ≥40% |
| | or Hypotension requiring high dose or multiple vasopressors or Grade 3 organ toxicity or grade |
| | 4 transaminitis |
| Grade 4 | Life-threatening symptoms - Requirement for ventilator support or Grade 4 organ toxicity |
| | (excluding transaminitis) |
| Grade 5 | Death |

Grades 2-4 refer to CTCAE v4.0 grading.

### 10.1 Definitions

The following definitions are based on the Code of Federal Regulations Title 21 Part 312.32 (21CFR312.32(a)).

**Adverse Event:** Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

**Suspected Adverse Reaction:** Any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of IND safety reporting, "reasonable possibility" means there is evidence to suggest a causal relationship between the drug and the adverse event. Suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

Life-Threatening Adverse Event Or Life-Threatening Suspected Adverse Reaction: An adverse event or suspected adverse reaction is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an

adverse event or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

**Serious Adverse Event or Serious Suspected Adverse Reaction:** An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes:

- Death
- A life-threatening adverse event
- Inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- A congenital anomaly/birth defect
- An important medical event

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition

If either the IND sponsor or the investigator believes the event is life-threatening or serious, the event must be evaluated by the sponsor for expedited reporting (21CRF 312.32(a)).

Unexpected adverse event or unexpected suspected adverse reaction: An adverse event or suspected adverse reaction is considered "unexpected" if it is not listed in the investigator brochure or is not listed at the specificity or severity that has been observed; or, if an investigator brochure is not required or available, is not consistent with the risk information described in the general investigational plan or elsewhere in the current application, as amended.

**Expedited (Rapid) Reporting:** Certain events may require rapid notification to entities providing patient safety oversight (e.g. IRB) as detailed in Section 10.5.

The categories for AE attribution to study treatment are as follows:

- Definite clearly related
- Probable likely related
- Possible may be related
- Unlikely doubtfully related
- Unrelated clearly not related

The following definitions are from the Masonic Cancer Center's Standard Operating Procedure (SOP) Deviation Reporting:

<u>Major Deviation:</u> A deviation or violation that impacts the risks and benefits of the research; may impact subject safety, affect the integrity of research data and/or affect a subject's willingness to participate in the research. Deviations that place a subject at risk, but do not result in harm are considered to be major deviations.

<u>Minor Deviation</u>: A deviation or violation that does not impact subject safety, compromise the integrity of research data and/or affect a subject's willingness to participate in the research.

### **10.2 Event Documentation**

Event monitoring and documentation begins with the 1<sup>st</sup> dose of TriKEs.

For the purposes of this study, selected expected adverse events will be assessed using the Targeted Toxicity Worksheet (Appendix VI) and any unexpected events will be collected at the following time points in relation to the GTB-3550 TriKE infusions through Day 29:

- Prior to the infusion start of each 24 hour infusion (i.e. Day 1, 2, 3, 4, and Day 8, 9, 10, 11, and Day 15, 16, 17, 18)
- At the end of the final infusion of each block (i.e. Day 5, Day 12, Day 19)
- Day 22
- Day 29

At each time point, the worst grade of the targeted toxicity since the last assessment or the previous 24 hours (whichever is shorter) will be recorded in addition to any unexpected toxicities felt at least possibly related the study treatment.

If a patient discontinues study therapy early or otherwise does not receive treatment as planned, the targeted toxicity assessment time points may be adjusted or eliminated; however, patients must be assessed for a minimum of 28 days from the 1<sup>st</sup> dose of study drug.

If a patient is not abiding by the standard of care study calendar (Section 8.1), collection of the corresponding targeted events (and research related samples) also may be altered or discontinued on an individual patient basis, as appropriate.

Monitoring for adverse events will end after the last targeted assessment; however, the investigator is obligated, upon knowledge of, to report any event meeting the criteria in Section 10.5.

# 10.3 Dose Limiting Toxicity Documentation and Reporting (Phase I Dose Finding)

The following events count toward dose limiting toxicity (DLT) during the Phase I dose finding component and must be reported the UMN Multisite Program Manager per Section 10.6.

Note: DLT events are only reported for patients enrolled in the Phase I portion of the trial; however, any patient experiencing a DLT is not eligible to continue treatment per Section 7.5.

A DLT is defined as a related treatment emergent toxicity that occurs within 28 days after the 1<sup>st</sup> TriKE dose with the exception of those that are clearly and incontrovertibly due to extraneous causes:

- Any Grade 4 or 5 non-hematologic events
- Grade 3 non-hematologic adverse events lasting more than 72 hours, **except** the following:
  - Non-sustained (< 7 days) Grade 3 liver function tests (ALT/AST, alkaline phosphatase, total or direct bilirubin) abnormalities in the absence of clinical signs of hepatic dysfunction (lethargy, confusion, anorexia, pruritus or tremors).
  - Non-sustained Grade 3 QTc prolongation (< 72 hours) in the absence of cardiac arrhythmia
  - Grade 3 electrolyte disturbances that resolve, with or without intervention, to
     Grade 2 levels within 72 hours
  - Grade 3 fatigue
  - o Grade 3 anorexia
  - Grade 3 fever
  - Grade 3 infection
- Hematologic Toxicity Given that AML and MDS inherently leads to low neutrophils and platelets, standard grading cannot be used as many of these patients technically meet criteria for "grade 4" neutropenia or thrombocytopenia at baseline. Thus, the hematologic DLTs are listed below:
  - o AML
    - Grade 4 neutrophil count (< 500/µL) lasting ≥ 29 days from start of cycle in absence of evidence of active leukemia

- Grade 4 platelet count (< 25,000/µL) lasting ≥ 29 days from start of cycle in absence of evidence of active leukemia
- Any clinically significant bleeding that is not controllable with transfusion support

### MDS/mast cell diseases:

- Grade 4 neutrophil count (<500/µL) lasting ≥ 29 days from start of cycle in absence of evidence of active MDS/mast cell disease
- Grade 4 platelet count (<25,000/µL) lasting ≥ 29 days from start of cycle in the absence of active MDS/Mast cell disease
- Any clinically significant bleeding that is not controllable with transfusion support
- Grade 4 anemia, unexplained by the underlying disease
- Grade 3 infusion related, treatment related reaction including cytokine release syndrome which does not resolve within 72 hours despite best medical management (refer to Section 10 for modified CRS grading)
- Grade 3 or 4 Tumor Lysis Syndrome that does not resolve within 7 days with or without intervention
- Inability to complete at least one block of three 24 hour infusions due to any treatment emergent, treatment related toxicity.

# 10.4 Early Study Stopping Rules - Event Documentation and Reporting (Phase II Dose Expansion)

Early study stopping rules for the Phase II dose expansion component patients are:

- Grade 4-5 non-hematologic, non-relapse, non-infectious toxicity (except fever) by 42 days after the start of the first GTB-3550 TriKE treatment block
- Non-relapse, non-infectious treatment related mortality (TRM) within 60 days of starting GTB-3550 TriKE treatment

Meeting either stopping rule criterion temporarily will halt study enrollment until the event is fully evaluated and the Principal Investigator and GT Biopharma make a decision regarding the continuation of the trial. Any patients currently receiving treatment may continue after discussion with the study PI and GT Biopharma.

Events that count toward dose limiting toxicity and early stopping rules do not necessarily constitute a serious adverse event requiring expedited reporting and should be reported as such only if they meet the criteria for expedited reporting as defined in Section 10.6.

### 10.5 Documentation of Death and Reporting Requirements

Deaths during treatment and the follow-up period, including death due to disease, will be recorded as an SAE and reported per Section 10.6. Deaths due to disease should be recorded as a Grade 5 Neoplasm.

In addition, even after the follow-up period ends, the death date must be documented in the patient follow-up tab in upon knowledge using the comment field in survival status section to record the cause.

June 4, 2021 

### 10.6 Participating Sites Event Reporting Table

| Event Type | Reporting Timeframe | Form to Use | Email to |
|---|---|---|---|
| Any event meeting the | Within 24 hours of | Paper SAE Report Form | Masonic Cancer Center (MCC) |
| definition of serious | knowledge | | Multisite Program Manager |
| Dose Limiting Toxicity | Within 24 hours of | DLT Event Form | |
| Event | knowledge | | |
| Stopping Rule Event | Within 24 hours of | Stopping Rule Event | |
| | knowledge | Form | |
| Major Deviations, as | Within 5 working days of | Record in Deviations | |
| defined in Section 10.1. | knowledge | Tab, generate report and | |
| | | have PI sign | |
| Minor Deviations, as | Reporting not applicable | Record in Deviations | Not applicable |
| defined in Section 10.1. | | Tab – signed report not | |
| | | required | |

Participating Sites are responsible for reporting to Local institutional IRB or other entities per institutional policies and guidelines.

The Multisite Program Manager will forward all reports to GT Biopharma and within 3 business hours.

GT Biopharma/ is responsible for submission of IND safety reports to the FDA per federal regulations.

# 10.7 UMN Required Reporting: UMN IRB, GT Biopharma, and Masonic Cancer Center's SAE Coordinator

| Entity<br>Reported To: | Criteria for reporting | Timeframe | Form to Use | Report to |
|---|---|---|---|---|
| U OF MN IRB | Information that indicates a new or increased risk, or safety issue. Unexpected Death per UMN requirements. Clinical deviations per current IRB reporting requirements (UMN patients only) | 5 business<br>days | Ethos Reportable New Information (RNI) Deviation Report and | Via with copy GT Biopharma* |
| GT<br>Biopharma<br>and ** | Any event meeting the definition of serious regardless of attribution Events that count toward dose limiting toxicity during the dose finding component or an early study stopping rule during the expanded component | Within 24 hours<br>of knowledge<br>At time of<br>reporting | CTO SAE Report<br>Form<br>Appropriate form | GT Biopharma and |

<sup>\*</sup>GT Biopharma/ is responsible for submission of IND safety reports to the FDA per federal regulations.

### 11 Study Data Collection and Monitoring

### 11.1 Data Management

| | This study will collect regulatory and clinical data using |
|---|---|
| | The database resides on dedicated secure and PHI compliant hardware consisting of 3 physical servers: dev, DR, and production. All the data servers are managed by the all procedures related for PHI compliant servers (as required by the Center of Excellence for HIPAA Data) apply to databases. |
| | The integrated data will be stored in PHI compliant servers managed by with access given to those authorized users in the Clinical and Translation Science Institute Informatics team (CTSI BPIC and MCC CISS). |
| | Key study personnel are trained on the use of and will comply with protocol specific instructions embedded within the . |
| 11. | 2 Case Report Forms |
| | Participant data will be collected using protocol specific electronic case report forms (e-CRF) developed based on its library of standardized forms. The e-CRFs will be approved by the lead center PI and the UMN biostatistician prior to release for use. The Study Coordinator or designee will be responsible for registering the patient into at time of study entry, completing e-CRF based on the patient specific calendar, and updating the patient record until patient death or end of required study participation. |
| 11. | 3 Data and Safety Monitoring |
| | The study will be in compliance with the |

June 4, 2021 

The site PI will comply with at least twice yearly monitoring of the project by their site's internal monitoring staff. Monitoring reports are forwarded to the U of MN Multisite Program Manager who will forward to the reports to GT Biopharma Refer to the Procedures Manual for Participating Sites for additional information.

All sites must permit study-related monitoring, audits, and inspections by the IND Sponsor (GT Biopharma and/or their designee), IRB, government regulatory bodies, and compliance groups. The investigator will make available all study related documents (e.g. source documents, regulatory documents, data collection instruments, study data, etc.). The investigator will ensure the capability for inspections of applicable study-related facilities (e.g. pharmacy, diagnostic laboratory, etc.) will be available for trial related monitoring, audits, or regulatory inspections.

### 11.4 UMN Led Teleconferences – Participating Sites, GT Biopharma



Regular teleconferences will be held to facilitate communication between the participating sites and IND sponsor/representative regarding the study's progress, including patient updates, a summary of safety reports, dose level/patient slot availability, case report form completion, and other issues for discussion. The Masonic Cancer Center Multisite Program Manager is responsible for arranging these teleconferences and preparing the agenda. Meetings occur every 2 weeks; however, they may be scheduled more or less frequently at the discretion of the lead institution. Participation of a minimum of one representative from each participating clinical site is expected. Attendance by

These teleconferences are in addition to other previously described site interactions including centralized patient registration, institutional and MCC required reporting of safety related issues, and case report form completion in the study's central database

### 11.5 Record Retention

The investigator will retain essential documents (e.g. study records including source data, copies of case report form, consent forms, HIPAA authorizations, and all study correspondence) until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents should be retained for a longer period

however if required by the applicable regulatory requirements or by an agreement with the sponsor.

It is the responsibility of the sponsor (GT Biopharma) to inform the investigator/institution as to when these documents no longer need to be retained.

### 12 Statistical Considerations

### 12.1 Study Design and Endpoints

This is a multisite Phase I/II study of GTB-3550 trispecific killer cell engager (TriKE) for the treatment of high risk MDS and relapsed AML. Once the MTD is identified, the objective will be to confirm safety and obtain preliminary estimates of efficacy as measured by the objective response, the **primary trial endpoint** as assessed between Day 21 and Day 42. For AML clinical response includes complete remission with or without hematologic or platelet recovery (CR, CRi or CRp) or partial response. For MDS clinical response includes complete remission, marrow CR (with incomplete peripheral blood count normalization), partial response or hematologic improvement (HI). For advanced systemic mastocytosis response is considered a decrease in mast cell burden in bone marrow or serum tryptase level by at least 30%.

All patients completing Block #1 will be evaluable for DLTs and toxicities. Patients who discontinue therapy prior to completion of both Block #1 and Block #2 will be replaced. Patients completing Block #1 and Block #2, but come off treatment for disease progression, will still be evaluable for efficacy and will not be replaced. If needed a subgroup of patients receiving all 3 blocks will also be evaluated for response as a secondary population. We expect that the number of patients coming off therapy after only completing block #1 will be minimal.

**Secondary trial endpoints** will include toxicity through Day 29 and overall survival (OS) at 6 months from 1<sup>st</sup> dose of study drug.

### Phase I component: Estimating the MTD of GTB-3550 TriKE:

The first phase is a dose finding study with the aim of establishing the MTD of GTB-3550 TriKE when given as a block of four 24 hour infusions with a 72 hour break for 3 consecutive weekly courses in patients with CD33-expressing high risk myelodysplastic syndromes, refractory/relapsed acute myeloid leukemia or advanced systemic mastocytosis. The MTD will be identified using the continual reassessment method (CRM)<sup>44</sup>.

The MTD will be defined as the dose that most closely corresponds to a dose limiting toxicity (DLT) rate of 20%. Dose limiting toxicity (DLT) is defined Section 7.2.1. Determination of the target rate of 20% was based on clinical input and acceptability.

Seven dose levels of GTB-3550 TriKE will be tested (5.0  $\mu$ g/kg, 10.0  $\mu$ g/kg, 25.0  $\mu$ g/kg; 50.0  $\mu$ g/kg, 100.0  $\mu$ g/kg, 150  $\mu$ g/kg, and 200  $\mu$ g/kg daily dose). The CRM uses a Bayesian framework that combines experience from patients in the earlier part of the trial with clinicians' initial best probability estimates of DLT at each dose. We are using a one parameter power model for the probability of DLT, where the probability at each dose i, is modeled as  $F(d, \alpha) = d_i e^{xp(\alpha)}$  where  $\alpha$  is distributed a priori as a normal random variable with mean 0 and variance 0.5. The variance of the prior distribution, 0.5, was determined through simulations to balance accuracy and patient safety.

**Revision 5/5/2021**: Seven dose levels of GTB-3550 TriKE are now being tested per 7.2.1 (5.0  $\mu$ g/kg, 10.0  $\mu$ g/kg, 25.0  $\mu$ g/kg, 50.0  $\mu$ g/kg, 100.0  $\mu$ g/kg, 150.0  $\mu$ g/kg and 200  $\mu$ g/kg daily dose) using an expected "true" probability of 17% for DLTs at 150.0  $\mu$ g/kg (median probability between 100 and 200  $\mu$ g/kg daily dose) and the same target DLT rate of 20%.

The prior mean for the probability of DLT for the six doses (i.e. the power model skeleton) are 3%, 5%, 7%, 10%, 14% and 20%, respectively. As the study progresses, updated probabilities of DLT are computed before each new cohort of patients is enrolled and both patients of each cohort have reached Day 28 (end of the DLT assessment period) prior to enrollment of a subsequent cohort. Each subsequent cohort will be assigned to the most appropriate dose based on these updated probabilities. Eventually the final dose (within our proposed sample of 30 patients) will be identified as the dose most closely associated with a DLT rate of 20%. To promote patient safety: 1) we will enroll cohorts of 2 patients starting at the 1st dose; and 2) dose levels will not be skipped when escalating.

# Phase II Extension: Studying the efficacy of GTB-3550 TriKE for the endpoint of objective response:

After completion of the dose finding trial, the final dose will be carried forward into an uncontrolled two-stage Phase II extension trial to confirm safety and make a preliminary determination of the activity level. For advanced MDS/AML, the lack of

defined effective alternative therapies precludes a control regimen for comparisons at this stage of testing. If the Phase I trial enrolls fewer than 14 patients at the MTD, we will employ a Simon's Minimax two-stage design<sup>45</sup> with the possibility to discontinue after the 1<sup>st</sup> stage if the response rate is low.

- Stage 1: Enroll a total of 13 patients (including all treated at the MTD in Phase
   I). If 3 or more of these respond, the trial will continue to stage 2.
- Stage 2: Enroll an additional 17 patients. If 10 of 30 patients respond, GTB-3550 TriKE will be considered promising for further investigation.

If the Phase I trial enrolls more than 13 patients at the MTD, we will adjust the futility rule above for the two-stage design with the given number of patients enrolled at the MTD.

### 12.2 Statistical Analysis

Response will be estimated with simple proportions and descriptive plots. The secondary endpoint of OS will be estimated with Kaplan-Meier curves. Safety measures will be described with frequencies and proportions.

The change in number, phenotype and function of NK cells from baseline to the end of treatment will be correlated with clinical response using appropriate regression analyses such as Cox or Logistic regression. Assessment of serum TriKE levels will be determined using descriptive statistics.

### 12.3 Sample Size Justification

### Trial Size Determination:

Assuming a target DLT probability of 20%, an effect size or odds ratio of 1.7 and a commonly used accuracy index of 0.5, the initial sample size is 27. We conservatively rounded to 30 patients.

Operating

characteristics for various 'true' probabilities are listed in Table 1.



If fewer than 14 patients are enrolled at the MTD, the Phase II extension trial using the Simon's two-stage design will require 30 patients to test the null hypothesis that the response rate is <20% versus the alternative that the response rate is ≥40% after assuming 80% power and a significance level of 0.05.

If the Phase I trial enrolls more than 13 patients at the MTD, we will adjust the futility rule of the two-stage design while maintaining the constraints of 80% power, a significance level of 0.05 and using a maximum of 30 patients. We will choose the rule that minimizes the expected sample size given a true response rate equivalent to the null hypothesis. We expect that approximately 44 patients will be required due to use of patients from the Phase I trial in the Phase II extension but the sample size may be as high as 57. Enrollment is expected to be 1-2 patients per month.

### 12.4 Monitoring Guidelines (Study Stopping Rule Events)

During the CRM, the trial will stop if the posterior probability that the lowest dose is more toxic than the target is greater than 90%.

After the MTD has been established stopping rules will also be employed to monitor excess toxicity outside of the Phase I trial<sup>47</sup>.

Meeting either stopping rule criteria temporarily will halt enrollment per Section 10.4.

- (1) Grade 4-5 non-hematologic, non-relapse, non-infectious toxicity (except fever) by 42 days after the start of the first GTB-3550 TriKE treatment block: We will construct a boundary such that the probability of early stopping is at most 10% if the toxicity rate is equal to 10%. Assuming 27 additional patients are enrolled after phase I, the upper stopping boundary for toxicity would be 2/3, 3/8, 4/13, 5/20, 6/26 or 7 events.
- (2) **Non-relapse, non-infectious treatment related mortality** within 60 days of starting GTB-3550 TriKE treatment: Assuming the same parameters as in (1), the upper stopping boundary for TRM will be 2/3, 3/8, 4/13, 5/20, 6/26 or 7 events. If the true rates of both toxicity and TRM are 30%, the probability of early stopping will be 88% for each guideline.

### 13 Conduct of the Study

### 13.1 Good Clinical Practice

The study will be conducted in accordance with the appropriate regulatory requirement(s). Essential clinical documents will be maintained to demonstrate the validity of the study and the integrity of the data collected. Master files should be established at the beginning of the study, maintained for the duration of the study and retained according to the appropriate regulations.

### 13.2 Ethical Considerations

The study will be conducted in accordance with ethical principles founded in the Declaration of Helsinki. The IRB will review all appropriate study documentation in order to safeguard the rights, safety and well-being of the patients. The study will only be conducted at sites where IRB approval has been obtained. The protocol, consent, written information given to the patients, safety updates, annual progress reports, and any revisions to these documents will be provided to the IRB by the investigator.

### 13.3 Informed Consent

All potential study participants will be given a copy of the IRB-approved consent to review. The investigator or designee will explain all aspects of the study in lay language and answer all questions regarding the study. If the participant decides to participate in the study, he/she will be asked to sign and date the consent document. Patients who refuse to participate or who withdraw from the study will be treated without prejudice.

### 14 References

- 1. Taylor PR, Reid MM, Stark AN, Bown N, Hamilton PJ, Proctor SJ. De novo acute myeloid leukaemia in patients over 55-years-old: a population-based study of incidence, treatment and outcome. Northern Region Haematology Group. *Leukemia*. 1995;9(2):231-237.
- 2. Ostgard LS, Kjeldsen E, Holm MS, et al. Reasons for treating secondary AML as de novo AML. *Eur J Haematol*. 2010;85(3):217-226.
- 3. Vardiman JW, Thiele J, Arber DA, et al. The 2008 revision of the World Health Organization (WHO) classification of myeloid neoplasms and acute leukemia: rationale and important changes. *Blood*. 2009;114(5):937-951.
- 4. Mufti GJ, Bennett JM, Goasguen J, et al. Diagnosis and classification of myelodysplastic syndrome: International Working Group on Morphology of myelodysplastic syndrome (IWGM-MDS) consensus proposals for the definition and enumeration of myeloblasts and ring sideroblasts. *Haematologica*. 2008;93(11):1712-1717.
- 5. Masters GA, Krilov L, Bailey HH, et al. Clinical cancer advances 2015: Annual report on progress against cancer from the American Society of Clinical Oncology. *J Clin Oncol*. 2015;33(7):786-809.
- 6. Caruana I, Diaconu I, Dotti G. From monoclonal antibodies to chimeric antigen receptors for the treatment of human malignancies. *Semin Oncol.* 2014;41(5):661-666.
- 7. Hermanson DL, Kaufman DS. Utilizing chimeric antigen receptors to direct natural killer cell activity. *Front Immunol*. 2015;6:195.
- 8. Glienke W, Esser R, Priesner C, et al. Advantages and applications of CAR-expressing natural killer cells. *Front Pharmacol.* 2015;6:21.
- 9. Vivier E, Raulet DH, Moretta A, et al. Innate or adaptive immunity? The example of natural killer cells. *Science*. 2011;331(6013):44-49.
- 10. Velardi A. Natural killer cell alloreactivity 10 years later. *Curr Opin Hematol*. 2012;19(6):421-426.
- 11. Anegon I, Cuturi MC, Trinchieri G, Perussia B. Interaction of Fc receptor (CD16) ligands induces transcription of interleukin 2 receptor (CD25) and lymphokine genes and expression of their products in human natural killer cells. *J Exp Med*. 1988;167(2):452-472.
- 12. Ravetch JV, Bolland S. IgG Fc receptors. Annu Rev Immunol. 2001;19:275-290.
- 13. Selvaraj P, Carpen O, Hibbs ML, Springer TA. Natural killer cell and granulocyte Fc gamma receptor III (CD16) differ in membrane anchor and signal transduction. *J Immunol*. 1989;143(10):3283-3288.
- 14. Perussia B, Ravetch JV. Fc gamma RIII (CD16) on human macrophages is a functional product of the Fc gamma RIII-2 gene. *Eur J Immunol*. 1991;21(2):425-429.
- 15. Klaassen RJ, Ouwehand WH, Huizinga TW, Engelfriet CP, von dem Borne AE. The Fcreceptor III of cultured human monocytes. Structural similarity with FcRIII of natural killer cells and role in the extracellular lysis of sensitized erythrocytes. *J Immunol*. 1990;144(2):599-606.
- 16. Nishikiori N, Koyama M, Kikuchi T, et al. Membrane-spanning Fc gamma receptor III isoform expressed on human placental trophoblasts. *Am J Reprod Immunol*. 1993;29(1):17-25.
- 17. Ravetch JV, Perussia B. Alternative membrane forms of Fc gamma RIII(CD16) on human natural killer cells and neutrophils. Cell type-specific expression of two genes that differ in single nucleotide substitutions. *J Exp Med*. 1989;170(2):481-497.
- 18. Lanier LL, Ruitenberg JJ, Phillips JH. Functional and biochemical analysis of CD16 antigen on natural killer cells and granulocytes. *J Immunol*. 1988;141(10):3478-3485.
- 19. Wirthmueller U, Kurosaki T, Murakami MS, Ravetch JV. Signal transduction by Fc gamma RIII (CD16) is mediated through the gamma chain. *J Exp Med*. 1992;175(5):1381-1390.
- 20. Cooper MA, Fehniger TA, Caligiuri MA. The biology of human natural killer-cell subsets. *Trends Immunol*. 2001;22(11):633-640.

- 21. Beziat V, Duffy D, Quoc SN, et al. CD56brightCD16+ NK cells: a functional intermediate stage of NK cell differentiation. *J Immunol*. 2011;186(12):6753-6761.
- 22. Vivier E, Nunes JA, Vely F. Natural killer cell signaling pathways. *Science*. 2004;306(5701):1517-1519.
- 23. Vivier E, Morin P, O'Brien C, Druker B, Schlossman SF, Anderson P. Tyrosine phosphorylation of the Fc gamma RIII(CD16): zeta complex in human natural killer cells. Induction by antibody-dependent cytotoxicity but not by natural killing. *J Immunol*. 1991;146(1):206-210.
- 24. Nimmerjahn F, Ravetch JV. Fcgamma receptors as regulators of immune responses. *Nat Rev Immunol.* 2008;8(1):34-47.
- 25. Bryceson YT, Ljunggren HG, Long EO. Minimal requirement for induction of natural cytotoxicity and intersection of activation signals by inhibitory receptors. *Blood*. 2009;114(13):2657-2666.
- 26. Shore SL, Nahmias AJ, Starr SE, Wood PA, McFarlin DE. Detection of cell-dependent cytotoxic antibody to cells infected with herpes simplex virus. *Nature*. 1974;251(5473):350-352.
- 27. Laszlo A, Petri I, Ilyes M. Antibody dependent cellular cytotoxicity (ADCC)-reaction and an in vitro steroid sensitivity test of peripheral lymphocytes in children with malignant haematological and autoimmune diseases. *Acta Paediatr Hung.* 1986;27(1):23-29.
- 28. Natsume A, Niwa R, Satoh M. Improving effector functions of antibodies for cancer treatment: Enhancing ADCC and CDC. *Drug Des Devel Ther*. 2009;3:7-16.
- 29. Albertini MR, Hank JA, Sondel PM. Native and genetically engineered anti-disialoganglioside monoclonal antibody treatment of melanoma. *Cancer Chemother Biol Response Modif.* 2005;22:789-797.
- 30. Garcia-Foncillas J, Diaz-Rubio E. Progress in metastatic colorectal cancer: growing role of cetuximab to optimize clinical outcome. *Clin Transl Oncol*. 2010;12(8):533-542.
- 31. Garnock-Jones KP, Keating GM, Scott LJ. Trastuzumab: A review of its use as adjuvant treatment in human epidermal growth factor receptor 2 (HER2)-positive early breast cancer. *Drugs*. 2010;70(2):215-239.
- 32. Navid F, Santana VM, Barfield RC. Anti-GD2 antibody therapy for GD2-expressing tumors. *Curr Cancer Drug Targets*. 2010;10(2):200-209.
- 33. Winter MC, Hancock BW. Ten years of rituximab in NHL. *Expert Opin Drug Saf.* 2009;8(2):223-235.
- 34. Congy-Jolivet N, Bolzec A, Ternant D, Ohresser M, Watier H, Thibault G. Fc gamma RIIIa expression is not increased on natural killer cells expressing the Fc gamma RIIIa-158V allotype. *Cancer Res.* 2008;68(4):976-980.
- 35. Moore GL, Bautista C, Pong E, et al. A novel bispecific antibody format enables simultaneous bivalent and monovalent co-engagement of distinct target antigens. *MAbs.* 2011;3(6):546-557.
- 36. Preithner S, Elm S, Lippold S, et al. High concentrations of therapeutic IgG1 antibodies are needed to compensate for inhibition of antibody-dependent cellular cytotoxicity by excess endogenous immunoglobulin G. *Mol Immunol*. 2006;43(8):1183-1193.
- 37. Baselga J, Albanell J. Mechanism of action of anti-HER2 monoclonal antibodies. *Ann Oncol*. 2001;12 Suppl 1:S35-41.
- 38. Berinstein NL, Grillo-Lopez AJ, White CA, et al. Association of serum Rituximab (IDEC-C2B8) concentration and anti-tumor response in the treatment of recurrent low-grade or follicular non-Hodgkin's lymphoma. *Ann Oncol.* 1998;9(9):995-1001.
- 39. Holliger P, Hudson PJ. Engineered antibody fragments and the rise of single domains. *Nat Biotechnol.* 2005;23(9):1126-1136.
- 40. Chames P, Van Regenmortel M, Weiss E, Baty D. Therapeutic antibodies: successes, limitations and hopes for the future. *Br J Pharmacol*. 2009;157(2):220-233.

- 41. Scott AM, Wolchok JD, Old LJ. Antibody therapy of cancer. *Nat Rev Cancer*. 2012;12(4):278-287.
- 42. Vallera DA, Felices M, McElmurry D. IL15 Trispecific Killer Engagers (TriKE) Make Natural Killer Cells Specific to CD33b Targets While Also Inducing Persistence, In Vivo Expansion, and Enhanced Function. Clin Cancer Res; 22(14) July 15, 2016.
- 43. Lee DW, Gardner R, Porter DL, et al. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014;124(2):188-195.
- 44. O'Quigley J, Pepe M, Fisher L. Continual reassessment method: a practical design for phase 1 clinical trials in cancer. *Biometrics*. 1990;46(1):33-48.
- 45. Simon R. Optimal two-stage designs for phase II clinical trials. *Control Clin Trials*. 1989;10(1):1-10.
- 46. Cheung YK. Sample size formulae for the Bayesian continual reassessment method. *Clin Trials*. 2013;10(6):852-861.
- 47. Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. *Biometrics*. 2005;61(2):540-545.

June 4, 2021 

### **Appendix I - Karnofsky Performance Status**

| | Karnofsky Performance Scale |
|---|---|
| Percent | Description |
| 100 | Normal, no complaints, no evidence of disease. |
| 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| 80 | Normal activity with effort; some signs or symptoms of disease. |
| 70 | Cares for self, unable to carry on normal activity or to do active work. |
| 60 | Requires occasional assistance, but is able to care for most of his/her needs. |
| 50 | Requires considerable assistance and frequent medical care. |
| 40 | Disabled, requires special care and assistance. |
| 30 | Severely disabled, hospitalization indicated. Death not imminent. |
| 20 | Very sick, hospitalization indicated. Death not imminent. |
| 10 | Moribund, fatal processes progressing rapidly. |
| 0 | Dead. |

# Appendix II - Revised International Prognostic Scoring System (IPSS-R) for Myelodysplastic Syndromes and Risk Assessment Calculator Link

Developed by the International Working Group for the Prognosis of MDS (IWG-PM) under the aegis of the MDS Foundation, Inc.

https://www.mds-foundation.org/ipss-r-calculator/

### IPSS-R Cytogenetic Risk Groups\*,\*\*

| Cytogenetic prognostic subgroups | Cytogenetic abnormalities |
|---|---|
| Very good | -Y, del(11q) |
| Good | Normal, del(5q), del(12p), del(20q), double including del(5q) |
| Intermediate | del(7q), +8, +19, i(17q), any other single or double independent clones |
| Poor | -7, inv(3)/t(3q)/del(3q), double including -7/del(7q), Complex: 3 abnormalities |
| Very poor | Complex: >3 abnormalities |

### **IPSS-R Prognostic Score Values\***

| Prognostic<br>variable | 0 | 0.5 | 1 | 1.5 | 2 | 3 | 4 |
|---|---|---|---|---|---|---|---|
| Cytogenetics | Very<br>Good | | Good | | Intermediate | Poor | Very Poor |
| BM Blast % | ≤2 | | >2-<br><5% | | 5-10% | >10% | |
| Hemoglobin | ≥10 | | 8-<10 | <8 | | | |
| Platelets | ≥100 | 50-<br><100 | <50 | | | | |
| ANC | ≥0.8 | <0.8 | | | | | |

June 4, 2021 

IPSS-R Prognostic Risk Categories/Scores\*

| RISK CATEGORY | RISK SCORE |
|---------------|------------|
| Very Low | ≤1.5 |
| Low | >1.5 - 3 |
| Intermediate | >3 - 4.5 |
| High | >4.5 - 6 |
| Very High | >6 |

<sup>\*</sup>Greenberg, Tuechler, Schanz et al, Revised International Prognostic Scoring System (IPSS-R) for Myelodysplastic Syndrome, Blood 120: 2454, 2012

June 4, 2021 

<sup>\*\*</sup>Schanz J et al, J Clin Oncology 2012; 30:820.

### **Appendix III - Response Criteria**

### **Acute Leukemias:**

- Morphologic complete remission (CR): ANC ≥ 1,000/mcl, platelet count ≥ 100,000/mcl, < 5% bone marrow blasts, no Auer rods, no evidence of extramedullary disease. (No requirements for marrow cellularity, hemoglobin concentration).
- Morphologic complete remission with incomplete platelet recovery (CRp): Same as CR platelet count < 100,000/mcl.</li>
- Morphologic complete remission with incomplete blood count recovery (CRi): Same as CR but ANC may be < 1,000/mcl and/or platelet count < 100,000/mcl.</li>
- Partial remission (PR): ANC ≥ 1,000/mcl, platelet count > 100,000/mcl, and at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts < 5% with persistent Auer rods.

### Myelodysplastic Syndromes (MDS):

| Category | Response criteria (responses must last at least 4 wk) |
|---|---|
| Complete | Bone marrow: ≤ 5% myeloblasts with normal maturation of all cell lines* |
| remission | Persistent dysplasia will be noted*† |
| | Peripheral blood‡ |
| | Hgb ≥ 11 g/dL |
| | <ul> <li>Platelets ≥ 100 x 10<sup>9</sup>/L</li> </ul> |
| | <ul> <li>Neutrophils ≥ 1.0 x 10<sup>9</sup>/L†</li> </ul> |
| | Blasts 0% |
| Partial remission | All CR criteria if abnormal before treatment except: |
| | <ul> <li>Bone marrow blasts decreased by ≥ 50% over pretreatment but still &gt; 5%</li> </ul> |
| | Cellularity and morphology not relevant |
| Marrow CR | Bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment† |
| | Peripheral blood: if HI responses, they will be noted in addition to marrow CR† |
| Stable disease | Failure to achieve at least PR, but no evidence of progression for ≥ 8 weeks |
| Cytogenetic | Complete |
| response | Disappearance of the chromosomal abnormality without appearance of new ones |
| | Partial |
| | At least 50% reduction of the chromosomal abnormality |
| Hematologic | Erythroid response (pretreatment,< 11 g/dL): |
| Improvement | Hgb increase by 1.5 g/dL Relevant reduction of units of RBC transfusions by an absolute |
| | number of at least 4 RBC transfusions/8 wk compared with the pretreatment transfusion |
| | number in the previous 8 wk. |
| | District reasons (pretractment < 100 V 100/L); |
| | Platelet response (pretreatment,< 100 X 109/L): Absolute increase of < 30 X 109/L for patients starting with 20 X 109/L platelets |
| | Increase from less than 20 X 109/L to greater than 20 X 109/L and by at least 100% |
| | Neutrophil response (pretreatment,< 1.0 X 109/L) At least 100% increase and an absolute increase 0.5109/L |
| | At least 100 /0 illolease and all absolute illolease0.3109/E |

MDS indicates myelodysplastic syndromes; Hgb, hemoglobin; CR, complete remission; HI, hematologic improvement; PR, partial remission; FAB, French-American-British; AML, acute myeloid leukemia; PFS, progression-free survival; DFS, disease-free survival. \*Dysplastic changes should consider the normal range of dysplastic changes (modification). †Modification to IWG response criteria.

‡In some circumstances, protocol therapy may require the initiation of further treatment (eg, consolidation, maintenance) before the 4-week period. Such patients can be included in the response category into which they fit at the time the therapy is started. Transient cytopenias during repeated chemotherapy courses should not be considered as interrupting durability of response, as long as they recover to the improved counts of the previous course.

Ref: Cheson BD, Greenberg DL, Bennett JM, et al. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 108: 419-425.

### Appendix IV - P450 Drug Interactions

### Flockhart Table ™

For complete table: http://medicine.iupui.edu/clinpharm/ddis/clinical-table accessed July 25, 2018

P450 Drug Interactions select substrates

Abbreviated "Clinically Relevant" Table

**SUBSTRATES** 

2D6 3A4,5,7

**Beta Blockers:** Macrolide antibiotics:

clarithromycin carvedilol

S-metoprolol erythromycin (not 3A5) NOT azithromycin propafenone timolol telithromycin

**Antidepressants:** Anti-arrhythmics:

amitriptyline quinidine→3-OH(not 3A5)

clomipramine

desipramine

Benzodiazepines: duloxetine alprazolam fluoxetine diazepam→3OH imipramine midazolam paroxetine

triazolam

Antipsychotics: Immune Modulators:

haloperidol cyclosporine

risperidone tacrolimus (FK506) thioridazine

sirolimus

Others:

**HIV Antivirals:** aripiprazole

indinavir atomoxetine ritonavir codeine saquinavir dextromethorphan nevirapine

doxepine flecainide

mexiletine Prokinetics: ondansetron cisapride

oxycodone

risperidone Antihistamines:

tamoxifen astemizole chlorpheniramine TAMOXIFEN GUIDE

tramadol

venlafaxine Calcium Channel Blockers:

> amlodipine diltiazem felodipine

June 4, 2021 

### **SUBSTRATES**

2D6 3A4,5,7

nifedipine nisoldipine nitrendipine verapamil

### **HMG CoA Reductase Inhibitors:**

atorvastatin lovastatin NOT pravastatin NOT rosuvastatin simvastatin

### PDE-5 Inhibitors:

sildenafil tadalafil vardenafil

### Others:

alfentanyl
aripiprazole
boceprevir
buspirone
carbamazepine
gleevec
haloperidol
pimozide
quinine
tamoxifen
telaprevir

trazodone vincristine

June 4, 2021 

### **INHIBITORS**

- A Strong inhibitor is one that causes a > 5-fold increase in the plasma AUC values or more than 80% decrease in clearance.
- A Moderate inhibitor is one that causes a > 2-fold increase in the plasma AUC values or 50-80% decrease in clearance.
- A Weak inhibitor is one that causes a > 1.25-fold but < 2-fold increase in the plasma AUC values or 20-50% decrease in clearance.

2D6 3A4,5,7 **HIV Antivirals:** bupropion indinavir fluoxetine nelfinavir paroxetine ritonavir quinidine, clarithromycin **■** itraconazole ■ ketoconazole duloxetine nefazodone amiodarone erythromycin cimetidine grapefruit juice ■ verapamil₂ aripiprazole diphenhydramine suboxone chlorpheniramine diltiazem clomipramine doxepin cimetidine haloperidol amiodarone methadone NOT azithromycin ritonavir fluvoxamine terbinafine troleandomycin voriconazole

### **INHIBITORS**

- A Strong inhibitor is one that causes a > 5-fold increase in the plasma AUC values or more than 80% decrease in clearance.
- A Moderate inhibitor is one that causes a > 2-fold increase in the plasma AUC values or 50-80% decrease in clearance.
- A Weak inhibitor is one that causes a > 1.25-fold but < 2-fold increase in the plasma AUC values or 20-50% decrease in clearance.



| INDUCERS | |
|---|---|
| 2D6 | 3A4,5,7 |
| | carbamazepine efavirenz nevirapine phenobarbital phenytoin pioglitazone rifabutin rifampin St. John's Wort troglitazone |

Metabolizer Phenotypes:

PM = Poor

IM = Intermediate

EM = Extensive

UM = Ultrarapid

The Flockhart Table™ is © 2016 by The Trustees of Indiana University. All rights reserved.

June 4, 2021 

### Appendix V - Combined List of Drugs That Prolong QT/QTc

### CredibleMeds Filtered QTDrug List

CREDIBLEMEDS<sup>TM</sup>
powered by AZCERT.ORG

The last revision date: May 20, 2018

See Note below for safe use of this

**Table** 

Highlighted Drugs are those frequently used in

cancer patient care.

The drug list below contains drugs from the categories: Known Risk of TdP And Avoid in congenital long QT

| Generic Name | Brand Names<br>(Partial List) | Drug Class | Therapeutic Use | Risk<br>Category | Route |
|---|---|---|---|---|---|
| Aclarubicin (Only<br>on Non US<br>Market) | Aclacin, Aclacinomycine, Aclacinon, Aclaplastin, Jaclacin | Anti-cancer | Cancer | Risk of TdP<br>And Avoid in<br>congenital long<br>QT | injection |
| Amiodarone | Cordarone,<br>Pacerone,<br>Nexterone | Antiarrhythmic | Arrhythmia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Anagrelide | Agrylin, Xagrid | Phosphodiester ase 3 inhibitor | Thrombocythemia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Arsenic trioxide | Trisenox | Anti-cancer | Cancer (leukemia) | Risk of TdP And<br>Avoid in congenital<br>long QT | injection |
| Astemizole<br>(Removed from<br>Market) | Hismanal | Antihistamine | Allergic rhinitis | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Azithromycin | Zithromax, Zmax | Antibiotic | Bacterial infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Bepridil<br>(Removed from<br>Market) | Vascor | Antianginal | Angina Pectoris<br>(heart pain) | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Chloroquine | Aralen | Antimalarial | Malaria | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Chlorpromazine | Thorazine,<br>Largactil,<br>Megaphen | Antipsychotic /<br>Antiemetic | Schizophrenia,<br>nausea, many<br>others | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection,<br>suppositor<br>y |
| Cilostazol | Pletal | Phosphodiester ase 3 inhibitor | Intermittent claudication | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |

| Generic Name | Brand Names<br>(Partial List) | Drug Class | Therapeutic Use | Risk<br>Category | Route |
|---|---|---|---|---|---|
| Ciprofloxacin | Cipro, Cipro-XR,<br>Neofloxin | Antibiotic | Bacterial infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Cisapride<br>(Removed<br>from Market) | Propulsid | GI stimulant | Increase GI<br>motility | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Citalopram | Celexa, Cipramil | Antidepressant,<br>SSRI | Depression | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Clarithromycin | Biaxin, Prevpac | Antibiotic | Bacterial infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>inhaled |
| Cocaine | Cocaine | Local anesthetic | Anesthesia<br>(topical) | Risk of TdP And<br>Avoid in congenital<br>long QT | oral, nasal |
| Disopyramide | Norpace | Antiarrhythmic | Arrhythmia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Dofetilide | Tikosyn | Antiarrhythmic | Arrhythmia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Domperidone<br>(Only on Non<br>US Market) | Motilium, Motillium,<br>Motinorm Costi,<br>Nomit | Antiemetic | Nausea, vomiting | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection,<br>suppositor |
| Donepezil | Aricept | Cholinest<br>erase<br>inhibitor | Dementia<br>(Alzheimer's<br>Disease) | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Dronedarone | Multaq | Antiarrhythmic | Arrhythmia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Droperidol | Inapsine,<br>Droleptan, Dridol,<br>Xomolix | Antipsychotic/<br>Antiemetic | Anesthesia<br>(adjunct), nausea | Risk of TdP And<br>Avoid in congenital<br>long QT | injection |
| Erythromycin | E.E.S., Robimycin, EMycin, Erymax, Ery- Tab, Eryc Ranbaxy, Erypar, Eryped, Erythrocin Stearate Filmtab, Erythrocot, E-Base, Erythroped, Ilosone, MY-E, Pediamycin, Abboticin, Abboticin- ES, Erycin, PCE Dispertab, Stiemycine, Acnasol, Tiloryth | Antibiotic | Bacterial infection, increase GI motility | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |

| Generic Name | Brand Names<br>(Partial List) | Drug Class | Therapeutic Use | Risk<br>Category | Route |
|---|---|---|---|---|---|
| Escitalopram | Cipralex, Lexapro,<br>Nexito, Anxiset-E<br>(India), Exodus<br>(Brazil), Esto (Israel),<br>Seroplex, Elicea,<br>Lexamil, Lexam,<br>Entact (Greece),<br>Losita (Bangladesh),<br>Reposil (Chile),<br>Animaxen<br>(Colombia), Esitalo<br>(Australia), Lexamil<br>(South Africa) | Antidepressant,<br>SSRI | Depression<br>(major), anxiety<br>disorders | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Flecainide | Tambocor,<br>Almarytm, Apocard,<br>Ecrinal, Flécaine | Antiarrhythmic | Arrhythmia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Fluconazole | Diflucan, Trican | Antifungal | Fungal infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Gatifloxacin<br>(Removed from<br>Market) | Tequin | Antibiotic | Bacterial infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Grepafloxacin<br>(Removed from<br>Market) | Raxar | Antibiotic | Bacterial infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Halofantrine<br>(Only on Non<br>US Market) | Halfan | Antimalarial | Malaria | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Haloperidol | Haldol (US & UK), Aloperidin, Bioperidolo, Brotopon, Dozic, Duraperidol (Germany), Einalon S, Eukystol, Halosten, Keselan, Linton, Peluces, Serenace, Serenase, Sigaperidol | Antipsychotic | Schizophrenia,<br>agitation | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Ibogaine (Only on<br>Non US Market) | None | Psychedelic | Narcotic addiction, unproven | Risk of TdP And<br>Avoid in<br>congenital long<br>QT | oral |
| Ibutilide | Corvert | Antiarrhythmic | Arrhythmia | Risk of TdP And<br>Avoid in congenital<br>long QT | injection |
| Levofloxacin | Levaquin, Tavanic | Antibiotic | Bacterial infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Levomepromazine<br>(methotrimeprazine)<br>(Only on Non US<br>Market) | Nosinan, Nozinan,<br>Levoprome | Antipsychotic | Schizophrenia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |

| Generic Name | Brand Names<br>(Partial List) | Drug Class | Therapeutic Use | Risk<br>Category | Route |
|---|---|---|---|---|---|
| Levomethadyl<br>acetate<br>(Removed from<br>Market) | Orlaam | Opiate | Narcotic<br>dependence | Risk of TdP And<br>Avoid in congenital<br>long QT | |
| Levosulpiride<br>(Only on Non<br>US Market) | Lesuride, Levazeo,<br>Enliva (with<br>rabeprazole) | Antipsychotic | Schizophrenia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Mesoridazine<br>(Removed from<br>Market) | Serentil | Antipsychotic | Schizophrenia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Methadone | Dolophine, Symoron,<br>Amidone,<br>Methadose,<br>Physeptone,<br>Heptadon | Opiate | Narcotic<br>dependence, pain | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Moxifloxacin | Avelox, Avalox,<br>Avelon | Antibiotic | Bacterial infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Ondansetron | Zofran, Anset,<br>Ondemet,<br>Zuplenz, Emetron,<br>Ondavell, Emeset,<br>Ondisolv,<br>Setronax | Antiemetic | Nausea, vomiting | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection,<br>suppositor<br>y |
| Oxaliplatin | Eloxatin | Anti-cancer | Cancer | Risk of TdP And<br>Avoid in congenital<br>long QT | injection |
| Papaverine HCI<br>(Intra-coronary) | none | Vasodilator,<br>Coronary | Diagnostic adjunct | Risk of TdP And<br>Avoid in congenital<br>long QT | injection |
| Pentamidine | Pentam | Antifungal | Fungal infection<br>(Pneumocystis<br>pneumonia) | Risk of TdP And<br>Avoid in congenital<br>long QT | injection,<br>inhaled |
| Pimozide | Orap | Antipsychotic | Tourette's Disorder | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Probucol<br>(Removed from<br>Market) | Lorelco | Antilipemic | Hypercholesterole mia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Procainamide | Pronestyl, Procan | Antiarrhythmic | Arrhythmia | Risk of TdP And<br>Avoid in congenital<br>long QT | injection |
| Propofol | Diprivan, Propoven | Anesthetic,<br>general | Anesthesia | Risk of TdP And<br>Avoid in congenital<br>long QT | injection |
| Quinidine | Quinaglute,<br>Duraquin, Quinact,<br>Quinidex, Cin-Quin,<br>Quinora | Antiarrhythmic | Arrhythmia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Roxithromycin<br>(Only on Non US<br>Market) | Rulide, Xthrocin,<br>Roxl-150, Roxo,<br>Surlid, Rulide,<br>Biaxsig, Roxar,<br>Roximycinv,<br>Roxomycin, Rulid, | Antibiotic | Bacterial infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |

| Generic Name | Brand Names<br>(Partial List) | Drug Class | Therapeutic Use | Risk<br>Category | Route |
|---|---|---|---|---|---|
| | Tirabicin,<br>Coroxin | | | | |
| Sevoflurane | Ultane, Sojourn | Anesthetic,<br>general | Anesthesia | Risk of TdP And<br>Avoid in congenital<br>long QT | inhaled |
| Sotalol | Betapace, Sotalex,<br>Sotacor | Antiarrhythmic | Arrhythmia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Sparfloxacin<br>(Removed from<br>Market) | Zagam | Antibiotic | Bacterial infection | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Sulpiride (Only<br>on Non US<br>Market) | Dogmatil,<br>Dolmatil, Eglonyl,<br>Espiride, Modal,<br>Sulpor | Antipsychotic,<br>atypical | Schizophrenia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>inhaled |
| Sultopride (Only<br>on Non US<br>Market) | Barnetil, Barnotil,<br>Topral | Antipsychotic,<br>atypical | Schizophrenia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral,<br>injection |
| Terfenadine<br>(Removed from<br>Market) | Seldane | Antihistamine | Allergic rhinitis | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Terlipressin (Only on Non US Market) | Teripress,<br>Glypressin, Terlipin,<br>Remestyp, Tresil,<br>Teriss and others | Vasoconstrictor | Septic shock | Risk of TdP And<br>Avoid in congenital<br>long QT | injection |
| Terodiline (Only<br>on Non US<br>Market) | Micturin, Mictrol (not bethanechol) | Muscle relaxant | Bladder spasm | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Thioridazine | Mellaril,<br>Novoridazine, Thioril | Antipsychotic | Schizophrenia | Risk of TdP And<br>Avoid in congenital<br>long QT | oral |
| Vandetanib | Caprelsa | Anti-cancer- | Cancer (thyroid) | Risk of TdP And<br>Avoid in congenital<br>long QT | |

Note: Medicines on this list are reviewed on an ongoing basis to assure that the available evidence supports their continued placement on this list. The list changes regularly and we recommend checking the website at crediblemeds.org for the most up-to-date information. There may be many additional brand names that are not listed on this form.

Disclaimer and Waiver: The information presented is intended solely for the purpose of providing general information about health-related matters. It is not intended for any other purpose, including but not limited to medical advice and/or treatment, nor is it intended to substitute for the users' relationships with their own health care providers. To that extent, by use of this website and the information it contains, the user affirms the understanding of the purpose and releases AZCERT, Inc. from any claims arising out of his/her use of the website and its lists. The absence of drugs from these lists should not be considered an indication that they are free of risk of QT prolongation or torsades de pointes. Many medicines have not been tested for this risk in patients, especially those with congenital long QT syndrome.

June 4, 2021 

### **Appendix VI - Targeted Expected Toxicities Worksheet**

| HM2015-39 | CTCAE v5 | Refer to Section 10.2 for time points |
|---|---|---|
| Patient Initials: | Date of Assessment: | Assessment Time Point: |

| Toxicity | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|
| Infusion related reaction | None | Mild transient reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interrup ion indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for ≤ 24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interrup ion of infusion); recurrence of symptoms following initial improvement; hospitalizatio indicated for clinical sequelae | Life-threatening consequences; urgent intervention indicated |
| Dyspnea | None or<br>no change | Shortness of breath wi h moderate exertion | Shortness of breath wi h minimal exer ion; limiting instrumental ADL | Shortness of breath at rest;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated |
| Hypoxia | None | | Decreased O <sub>2</sub> saturation with exercise (e.g., pulse oximeter < 88%) intermittent supplemental oxygen | Decreased oxygen saturation<br>at rest (e.g., pulse oximeter <<br>88% or PaO₂ ≤ 55 mm Hg) | Life-threatening airway<br>compromise; urgent<br>intervention indicated (e.g.,<br>tracheotomy or intubation) |
| Fever* | None | 38.0 - 39.0° C (100.4 -102.2° F) | > 39.0 - 40 0°C (102.3 - 104.0°F) | > 40.0 ∘ C (>104.0∘ F) for ≤ 24 hrs | > 40.0 ° C (>104.0° F) for > 24 hrs |
| Tachycardia* | None | Asymptomatic, interven ion not indicated | Non-urgent medical intervention indicated | Medical intervention or hospitalization indicated | Life-threatening and urgent intervention indicated |
| Chills | None | Mild sensation of cold; shivering; chattering of teeth | Moderate tremor of the entire body; narcotics indicated | Severe or prolonged, not responsive to narcotics | |
| Hypertension | None | Pre-hypertension (systolic BP<br>120 - 139 mm Hg or diastolic<br>BP 80 - 89 mm Hg) | Stage 1 hypertension (systolic BP 140 - 159 mm Hg or diastolic BP 90 - 99 mm Hg); medical intervention indicated; recurrent or persistent ≥ 24 hrs); symptomatic increase by >20 mm Hg (diastolic) or to >140/90 mm Hg if previously WNL; monotherapy indicated. | Stage 2 hypertension (systolic BP ≥ 160 mm Hg or diastolic BP ≥ 100 mm Hg); medical intervention indicated; more than one drug or more intensive therapy than previously used indicated. | Life-threatening consequences (e.g., malignant hypertension, transient or permanent neurologic deficit, hypertensive crisis); urgent intervention indicated. |
| Hypotension | None | Asymptomatic, interven ion not indicated | Non-urgent medical intervention indicated | Medical intervention or hospitalization indicated | Life-threatening and urgent intervention indicated |
| Edema | None | Localized to dependent areas,<br>no disability or functional<br>impairment | Moderate localized edema<br>and intervention indicated;<br>limi ing instrumental ADL | Severe localized edema and intervention indicated; limiting self care ADL | |
| Pneumonitis | None | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; oxygen indicated | Life-threatening respiratory<br>compromise; urgent<br>intervention indicated (e.g.<br>intuba ion or tracheotomy) |
| Headache | None | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | |
| Confusion<br>(Altered Mental<br>Status) | None | Mild disorientation | Moderate disorientation; limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening consequences; urgent intervention indicated |
| Rash | None | Covering < 10% body surface area (BSA) | Covering 10-30% body surface area (BSA) | >30% body surface area (BSA) | Generalized exfoliative, ulcera ive, or bullous dermatitis |
| Gait<br>Disturbance | None | Mild change in gait (eg, wide-<br>based, limping or hobbling) | Moderate change in gait (eg, wide-<br>based, limping or hobbling);<br>assistance device indicated;<br>limi ing instrumental ADL | Disabling; limiting self care ADL | |
| Ataxia<br>(Incoordination) | None | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; mechanical assistance indicated | |

\*refer to Section 7.1.2 - Monitoring for Signs of Immune Activation if present in a Phase I patient

| Person Completing Form: | ADL = activities of daily living |
|-------------------------|----------------------------------|

June 4, 2021 